#### The GlaxoSmithKline group of companies

| <b>Division</b> : Worldwide Development | Worldwide Development |
|---|---|
| Information Type | Reporting and Analysis Plan (RAP) |

| Title | : | A multicentre, randomised, double-blind (sponsor-unblinded), placebo-controlled, repeat dose study to investigate the safety and tolerability, pharmacokinetics, pharmacodynamics, and efficacy of GSK2982772 in subjects with active plaque-type psoriasis. |
|---|---|---|
| Compound Number | : | GSK2982772 |
| <b>Effective Date</b> | : | 24-May-2017 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 203167.
- This RAP is intended to describe the safety, tolerability, PK, PD, and efficacy analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | | 24-MAY-2017 |
|--------------|------------------------------------|--------------|
| Statistician | Statistician (Clinical Statistics) | |
| PPD | | 24-MAY-2017 |
| Manager Sta | ntistics (Clinical Statistics) | 24-MA 1-201/ |

## Approved by:

| PPD | | 24 MAY 2017 |
|---------------|------------------------------|-------------|
| Director Stat | istics (Clinical Statistics) | 24-MAY-2017 |

Copyright 2016 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## Clinical Study Identifier

#### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 5 |
| 2. | 2.1.<br>2.2. | Change:<br>Study O | KEY PROTOCOL INFORMATIONs to the Protocol Defined Statistical Analysis Planbjective(s) and Endpoint(s) | 7<br>7 |
| | 2.3.<br>2.4. | | esignal Hypotheses | |
| 3. | | | LYSES | |
| | 3.1.<br>3.2. | | Analysesalyses | |
| 4. | ANAL`<br>4.1. | | PULATIONS Deviations | |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 13 |
| 6. | STUD | | ATION ANALYSESw of Planned Analyses | |
| 7. | PRIMA<br>7.1. | ARY STA | TISTICAL ANALYSESnalysesOverview of Planned Efficacy Analyses | 16<br>16<br>16 |
| 8. | SECO<br>8.1. | | Pharmacokinetic Analyses Overview of Planned Pharmacokinetic Analyses Overview of Planned pharmacokinetic Analyses Drug Concentration Measures 8.1.3.1. Statistical Analysis of Pharmacokinetic Parameters | 19<br>19<br>19 |
| | 8.2. | 8.2.1.<br>8.2.2. | codynamic/Biomarker Analyses Overview of Planned Analyses Statistical Analysis of Inflammatory Biomarkers in the Skin Biopsy (Histopathological Scoring of Psoriatic Lesional Biopsies) | 20<br>20 |
| | | 8.2.3. | Statistical Analysis of mRNA from Skin Biopsies: Transcriptomic Data | |
| | 8.3. | Efficacy<br>8.3.1.<br>8.3.2. | AnalysesOverview of Planned Efficacy AnalysesStatistical Analysis of Efficacy Data | 22<br>22 |
| 9. | OTHE | R STATIS | STICAL ANALYSES2 | 24 |

| | | 011 51 | | Clinical Stud | |
|---|---|---|---|---|---|
| | 9.1. | | | ic Analyses | |
| | 9.1.1. | | of Planned Pharmacokinetic Analyses | | |
| | | 9.1.2. | | of Planned pharmacokinetic Analyses | |
| | | 9.1.3. | 9.1.3.1. | centration MeasuresStatistical Analysis of Pharmacokinetic | 24 |
| | | | | Parameters | 24 |
| | 9.2. | Explorato | ory Pharma | codynamic and Biomarker Analyses | 24 |
| | | 9.2.1. | | xploratory Biomarker Statistical Analyses | |
| | 9.3. | | | Analyses | |
| | | 9.3.1. | | xploratory Efficacy Statistical Analyses | |
| | 9.4. | Explorato | ory Pharma | codynamic / Efficacy Analyses | 29 |
| 10. | REFE | RENCES. | | | 30 |
| 11. | APPEI | NDICES | | | 31 |
| | 11.1. | | | Events | |
| | | | | efined Time & Events | |
| | 11.2. | | | ment Windows | |
| | | | | of Assessment Windows for Analyses | |
| | 11.3. | | | ent States and Phases | |
| | | 11.3.1. | | Phases | |
| | | 11.3.2. | | States | |
| | | | 11.3.2.1. | | |
| | 44.4 | A | | States for AE Data | |
| | 11.4. | Appendix 11.4.1. | ( 4: Data Di | splay Standards & Handling Conventions | ۵6 |
| | | 11.4.1. | | atment & Sub-group Display Descriptors | |
| | | 11.4.2. | | Baseline Definitions | |
| | | | 11.4.2.1. | | |
| | | | 11.7.2.2. | Data | 37 |
| | | 11.4.3. | Reporting | Process & Standards | |
| | 11.5. | | 5. Derived | I and Transformed Data | 40 |
| | | 11.5.1. | | | |
| | | 11.5.2. | | ulation | |
| | | 11.5.3. | | | |
| | | 11.5.4. | Pharmaco | kinetic | 41 |
| | | 11.5.5. | | | |
| | | 11.5.6. | Pharmaco | dynamic and Biomarker | 47 |
| | 11.6. | | | ure Withdrawals & Handling of Missing Data | |
| | | 11.6.1. | | : Withdrawals | |
| | | 11.6.2. | | of Missing Data | |
| | | | | Handling of Missing Dates | |
| | | | | Handling of Partial Dates | 49 |
| | | | 11.6.2.3. | Handling of Missing Data for Statistical | 40 |
| | 44 7 | ۸ | . <b>7</b> . \ /al | Analysis | 49 |
| | 11.7. | • • | | of Potential Clinical Importance | |
| | | 11.7.1.<br>11.7.2. | • | / Values | |
| | | 11.7.2.<br>11.7.3. | | | |
| | 11 8 | | | nter Studies | |

| | Clinical Study Ider | ntifier |
|---|---|---|
| | Appendix 9: Examination of Covariates, Subgroups & Other Strata | |
| | Appendix 10: Multiple Comparisons & Multiplicity | 55 |
| 11.11. | Appendix 11: Model Checking and Diagnostics for Statistical | |
| | Analyses | |
| | 11.11.1. Statistical Analysis Assumptions | 56 |
| 11.12. | Appendix 14 – Abbreviations & Trade Marks | 57 |
| | 11.12.1. Abbreviations | 57 |
| | 11.12.2. Trademarks | 58 |
| 11.13. | Appendix 15: List of Data Displays | 59 |
| | 11.13.1. Data Display Numbering | |
| | 11.13.2. Mock Example Shell Referencing | |
| | 11.13.3. Deliverable [Priority] | |
| | 11.13.4. Study Population Tables | |
| | 11.13.5. Safety Tables | |
| | 11.13.6. Safety Figures | 64 |
| | 11.13.7. Efficacy Tables | |
| | 11.13.8. Efficacy Figures | |
| | 11.13.9. Pharmacokinetic Tables | |
| | 11.13.10.Pharmacokinetic Figures | 72 |
| | 11.13.11. Pharmacodynamic and / or Biomarker Tables | |
| | 11.13.12. Pharmacodynamic (and / or Biomarker) Figures | |
| | 11.13.13.Biomarker / Efficacy Figures | |
| | 11.13.14.ICH Listings | |
| | 11.13.15.Non-ICH Listings | |
| 11.14. | Appendix 16: Example Mock Shells for Data Displays | |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This is the first study with GSK2982772 in subjects with active, plaque-type psoriasis. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamics (PD) and preliminary efficacy of GSK2982772. The intention of this study is to enable a fuller understanding of the mechanism of action and potential for clinical efficacy of GSK2982772 in PsO. |
| Protocol | This RAP is based on protocol amendment #2 [(Dated: 12/04/2017) of study GSK2982772 (GSK Document No. : 2015N251765_02)] and eCRF Version 3.0 |
| Primary<br>Objective | To investigate the safety and tolerability of 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 in subjects with active plaque-type psoriasis. |
| Primary<br>Endpoint | Safety and tolerability of GSK2982772 as assessed by clinical monitoring and reporting of adverse events, change in laboratory values, ECG, vital signs. |
| Study<br>Design | A multicentre, randomised, double-blind (sponsor-unblinded), placebo-controlled, repeat dose study proof of mechanism study. |
| | Approximately 30 subjects with active PsO will be randomised in a 2:1 ratio to GSK2982772 60mg BID and placebo respectively. |
| | Approximately 24 subjects with active PsO will be randomised in a 3:1 ratio to GSK2982772 60mg TID and placebo respectively |
| Planned | Safety and tolerability (primary). |
| Analyses | Pharmacokinetic (PK), Pharmacodynamic (PD) and clinical efficacy (secondary/exploratory). |
| Analysis | All subjects: all subjects screened for eligibility |
| Populations | Safety population: comprised all subjects who receive one dose of study treatment (placebo or GSK2982772). |
| | PK population: comprised subjects in the 'Safety' population for whom a pharmacokinetic sample was obtained and analysed. |
| Hypothesis | The primary objective of the study is to investigate the safety and tolerability of GSK2982772 60mg BID and 60mg TID following 12 weeks of treatment. No formal statistical hypotheses will be conducted to assess this objective. |
| | If appropriate, comparisons between the GSK2982772 60mg BID / 60mg TID arms and the placebo arm will be made to investigate the secondary inflammatory, mechanistic and efficacy objectives. Trends over time will be investigated for both treatment arms along with associations between each of the parameters. |
| Primary | Safety: |

Clinical Study Identifier

| Overview | Key Elements of the RAP |
|---|---|
| Analyses | <ul> <li>All data will be descriptively summarised, graphically presented and listed<br/>appropriately according to GSK's Integrated Data Standard Library (IDSL)<br/>standards.</li> </ul> |
| Secondary | General: |
| Analyses | <ul> <li>All data will be descriptively summarised, graphically presented and listed<br/>appropriately according to GSK's Integrated Data Standard Library (IDSL)<br/>standards.</li> </ul> |
| | <ul> <li>Modelling relationships between each of the mechanistic endpoints and<br/>also with the clinical endpoints using appropriate statistical modelling<br/>techniques to identify any trends.</li> </ul> |
| | <ul> <li>Trends over time will be investigated for all treatment arms along with<br/>associations between each of the key secondary and exploratory<br/>parameters.</li> </ul> |
| | <ul> <li>If appropriate, formal comparisons between each GSK2982772 arm and<br/>placebo will be made to investigate the secondary PD, mechanistic<br/>endpoints and efficacy.</li> </ul> |
| | Pharmacokinetic: |
| | No formal statistical analyses will be conducted. |
| | Pharmacodynamic/biomarker: |
| | <ul> <li>Descriptive statistics and/or graphical summaries for all PD and biomarker<br/>endpoints by treatment and time point.</li> </ul> |
| | Efficacy: |
| | <ul> <li>Descriptive statistics and/or graphical summaries of index lesion PLSS<br/>score by treatment and time point.</li> </ul> |
| | <ul> <li>(Percentage) change from baseline for the index lesion PLSS score will<br/>be analysed using repeated measures mixed effects model (MMRM),<br/>where appropriate.</li> </ul> |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 2 [(Dated: 12-Apr-2017)].

## 2.2. Study Objective(s) and Endpoint(s)

| Ob | Objectives | | Endpoints |
|---|---|---|---|
| Pri | Primary Objectives | | mary Endpoints |
| • | To investigate the safety and tolerability of 60 mg twice daily and 60 mg three times daily doses doses of GSK2982772 in subjects with active plaque-type psoriasis. | • | Adverse events Clinical laboratory values (clinical chemistry, haematology and urinalysis) Vital sign measurements (blood pressure, heart rate, respiratory rate and body temperature) 12-Lead ECG monitoring |
| Se | condary Objectives | Pri | mary Objectives |
| • | To investigate the pharmacokinetics of GSK2982772 in blood following 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 in subjects with active plaque-type psoriasis. | • | Pre-dose plasma concentrations of GSK2982772 at Days 43 (Week 6) and 85 (Week 12). Post-dose plasma concentrations of GSK2982772 on Days 1 and 43 (Week 6) at 1, 2, 4 and 6 hours post dose. |
| • | To investigate the effect of 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 on inflammatory biomarkers in skin biopsies from psoriatic skin lesions in subjects with active plaque-type psoriasis. | • | Change from baseline in histopathological scoring of psoriatic lesional biopsies which may include, but are not limited to the following as data permit: K16, CD3/CD11c, CD161, elastase positive dermal cells and epidermal thickness. mRNA expression of inflammatory gene transcripts which may include, but are not limited to the following as data permit: IL-4, IL-10, IL-17, IL-21, IL-22, IL-23, TNF and IFNγ on Days 1 (Week 0) and 43 (Week 6). |
| • | To investigate the effect of 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 on disease activity in subjects with active plaque-type psoriasis. | • | Percentage change from baseline and actual Psoriatic Lesion Severity Sum (PLSS) scores in the index lesion. |
| Ex | ploratory Objectives | Ex | ploratory Endpoints |
| • | To investigate the effect of 60 mg<br>twice daily doses and 60 mg three<br>times daily doses of GSK2982772<br>on disease activity in subjects with | • | Change from baseline in Psoriasis Area Severity Index (PASI) scores. The proportion of subjects who achieve PASI ≥ 50%, 75%, and 90% improvement from baseline score. |

Clinical Study Identifier

| - | | _ | Clinical Study Identifier |
|---|---|---|---|
| Obj | jectives | En | dpoints |
| | active plaque type psoriasis | • | Change from baseline and actual Physician Global Assessment (PGA). The proportion of subjects who achieve "clear" (0) or "almost clear" (1) on PGA. Change from baseline in body surface area (BSA). |
| • | To investigate the effect of 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 on inflammatory biomarkers in the blood of subjects with active plaque-type psoriasis. | • | Change from baseline in blood inflammatory markers which may include, but are not limited to the following as data permit: CRP, VEGF, S100A8, S100A9, IL-17, IL-22, and TNF. |
| • | To investigate the effect of 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 on transcriptome profiling of both blood and skin of subjects with active plaque-type psoriasis. | • | Transcriptomic analysis of mRNA isolated from blood and skin at Day 1 (Week 0) and Day 43 (Week 6). |
| • | To investigate pathway and target engagement following 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 in blood and skin biopsy tissue in subjects with active plaque-type psoriasis. | • | Pharmacology biomarker endpoints may include, but are not limited to the following Days 1 (Week 0), 43 (Week 6) and 85 (Week 12), as data permit: o Target Engagement Assay RIP1 (TEAR1) in blood and skin. o Total or phosprylated RIP1, MLKL, and RIP3, cleaved and total caspase 3 and caspase 8 signatures in skin. |
| • | To investigate the concentration of GSK2982772 in the skin of subjects with active plaque-type psoriasis after 60 mg twice daily doses of and 60 mg three times daily doses GSK2982772. | • | Pre-dose GSK2982772 concentrations in skin biopsies at Days 1 (Week 0) and 43 (Week 6), as data permit. |
| • | To investigate the effect of 60 mg twice daily doses and 60 mg three times daily doses of GSK2982772 on the patient reported outcomes (PROs) of subjects with active plaque-type psoriasis. | • | Change from baseline in Dermatology Life Quality Index (DLQI) score. Change from baseline and actual Visual Analogue Scale (VAS) itch score. |

#### 2.3. Study Design



| Overview of Study Design and Key Features | |
|---|---|
| Analysis | appropriate intervals by the GSK Safety Review Team (SRT). See SRT charter for further details. |
| | <ul> <li>The PLSS data will be reviewed in an unblinded manner when an appropriate number of subjects have completed Day 43. See the interim analysis chapter for further details.</li> <li>A formal interim analysis will be conducted after the completion of Cohort 1</li> </ul> |
| | and will only include those subjects randomised to a BID dosing regimen. |

## 2.4. Statistical Hypotheses

The primary objective of the study is to investigate the safety and tolerability of GSK2982772 60mg BID and 60mg TID following 12 weeks of treatment. No formal statistical hypotheses will be conducted to assess this objective.

If appropriate, comparisons between each GSK2982772 arm and the placebo arm will be made to investigate the secondary inflammatory, mechanistic and efficacy objectives. Trends over time will be investigated for both treatment arms along with associations between each of the parameters.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

In line with routine pharmacovigilance, an internal GSK Safety Review Team (SRT) which will include members of the 203167 study team, will review blinded safety data, including clinical laboratory parameters and adverse events, at appropriate intervals during the period of study conduct. Further details are outlined in the SRT charter.

In both cohorts, once an appropriate number of subjects randomised to GSK2982772 have completed Day 43 (Week 6), the PLSS data will be reviewed in an unblinded manner by a Data Review Committee (DRC) consisting of the GSK Project Physician Lead (PPL), the study statistician, the study pharmacokineticist, the Pattern Recognition Receptor (PRR) Discovery Performance Unit (DPU) Head, the Early Development Lead (EDL), the Safety Review Team (SRT) leader, or their designees on an ongoing basis. A physician external to the GSK2982772 project team may also be involved in the data review. Additional inflammatory biomarkers, clinical and mechanistic endpoints (e.g. target engagement) may be reviewed if available. No other member of the GSK core study team will be unblinded to this data. The primary purpose of these reviews will be to monitor PLSS changes for internal decision making purposes. A data review charter will identify the specific GSK individuals involved, outline in detail the activities of this review and how the integrity of the study will be maintained.

A formal interim analysis will be conducted after the completion of Cohort 1 and will only include those subjects randomised to a BID dosing regimen. The purpose of the

Clinical Study Identifier

interim analysis is primarily to provide the project team and key GSK stakeholders with an early indication of the safety and efficacy from the trial, and to facilitate decision making regarding the subsequent clinical development of GSK2982772.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. A completed subject is one who has completed all phases of the study including the follow-up visit.
- 3. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 4. All criteria for unblinding the randomisation codes have been met.
- 5. Randomisation codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All subjects | All subjects who were screened for eligibility. | Selected study population |
| Safety | <ul> <li>All subjects who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received<sup>[1]</sup></li> </ul> | <ul><li>Study population</li><li>Safety</li><li>Efficacy</li><li>PD</li></ul> |
| Pharmacokinetic | Subjects in the 'Safety' population for whom a pharmacokinetic sample was obtained and analysed. | • PK |

#### NOTES:

Please refer to Appendix 13: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

• Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

<sup>1.</sup> Any subjects who actually received both placebo and GSK2982772 due to dispensing errors will be assigned to GSK2982772, regardless of treatment duration

Clinical Study Identifier

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Time & Events |
| 11.2 | Appendix 2: Assessment Windows |
| 11.3 | Appendix 3: Treatment States and Phases |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |
| 11.8 | Appendix 8: Multicentre Studies |
| 11.9 | Appendix 9: Examination of Covariates, Subgroups & Other Strata |
| 11.10 | Appendix 10: Multiple Comparisons & Multiplicity |
| 11.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses. |
| 11.13 | Appendix 12: Abbreviations & Trade Marks |
| 11.14 | Appendix 13: Data Displays |
| 11.15 | Appendix 14: Example Mock Shells for Data Displays |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Randomisation | | | |
| Randomisation | | | Y |
| Subject Disposition | | | |
| Subject Disposition | Υ | | |
| Reasons for Screen Failure | Υ | | Y |
| Subjects by Centre | Υ | | |
| Reasons for Subject Withdrawal | | | Y |
| Subjects for Whom the Treatment Blind was Broken | | | Y |
| Planned and Actual Treatments | | | Y |
| Protocol Deviations | | | |
| Important Protocol Deviations | Υ | | Y |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Υ [1] |
| Populations Analysed | | | |
| Study Populations and Exclusions | Υ | | |
| Subjects Excluded from Any Population | | | Y |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Υ | | Y |
| PsO baseline characteristics – BSA,disease duration, prior treatments, naive phototherapy, PASI score, PLSS index lesions, PGA, Lesion severity area and score, history of tobacco use | Y | | Y |
| Race and Racial Combinations | Υ | | <b>Y</b> [2] |
| Prior and Concomitant Medications | | | |
| Current/Past Medical Conditions | Υ | | |
| Concomitant Medications | Y | | Y |
| Exposure and Treatment Compliance | | | |
| Exposure to Study Treatment | Υ | | Y |

#### NOTES:

- Y = Yes display generated.
- [1] Listing also includes analysis population exclusions.
- [2] Listing of race.

Clinical Study Identifier

#### 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Safety Analyses

## 7.1.1. Overview of Planned SafetyAnalyses

The primary safety analyses will be based on the "Safety" population, unless otherwise specified.

Table 3 provides an overview of the planned safety analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

Table 3 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | | Absol | ute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC | Υ | | Υ |
| Common (>=10%) AEs by Overall Frequency | Υ | Υ [1] | |
| All AEs by Maximum Intensity/Grade by SOC (and PT) | Υ | | |
| All Drug-Related AEs by SOC | Υ | | |
| Subjects & No. of Occurrences of Common Non-Serious AEs by SOC and PT | Υ | | |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Fatal Serious AEs | | | Υ |
| Non-Fatal Serious AEs | | | Υ |
| Serious AEs by SOC | Υ | | |
| Reasons for Considering as a Serious AE | | | Y |
| Drug-Related Serious AEs by SOC | Υ | | |
| AEs Leading to Withdrawal from Study / Permanent Discontinuation of Study | Υ | | Υ |
| Treatment by Overall Frequency | 1 | | Į. |
| Subjects and Number of Occurrences of Serious, Drug-Related Serious, Fatal | Υ | | |
| Serious, and Drug-Related Fatal Serious AEs | ' | | |
| Other Significant Adverse Events | | | Υ |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Plot of common AEs and relative risk will be generated.

#### 7.1.2. Overview of Clinical Laboratory Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Clinical Study Identifier

Table provides an overview of the planned analyses, with further details of data displays being presented in Appendix 1: List of Data Displays.

Table 5 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | | | | | |
| Chemistry Results | Υ | | | Υ | | |
| Emergent Chemistry Results by PCI Criteria | Υ | | | | | |
| Hematology | | | | | | |
| Hematology Results | Υ | | | Υ | | |
| Emergent Hematology Results by PCI Criteria | Υ | | | | | |
| Urinalysis | | _ | | | | |
| Urine Concentration | | | | Υ | | |
| Emergent Urinalysis Dipstick Results | Υ | | | | | |
| Hepatobiliary (Liver) | | _ | | | | |
| Liver Monitoring/Stopping Event Reporting | Υ | | | | | |
| Hepatobiliary Laboratory Abnormalities | Υ | | | | | |
| Medical Conditions for Subjects with Liver Stopping Events | | | Y | | | |
| Substance Use for Subjects with Liver Stopping Events | | | Y | | | |
| Scatter Plot of Maximum vs. Baseline for ALT | | Υ | | | | |
| Scatter Plot of Maximum ALT vs Maximum Total Bilirubin | | Υ | | | | |
| All Laboratory | | • | | | | |
| Laboratory Data for Subjects with Abnormalities of Potential Clinical Concern | | | Y | | | |
| Laboratory Data Abnormalities of Potential Clinical Importance | | | Y | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.3. Overview of Planned Other Safety Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Table provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

## Table 6 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Ch | ange | from BL |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumn | nary | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | | | | |
| Change from Baseline in ECG Values by Visit | | | | Υ | | |
| Maximum Change from Baseline in QTc Values by Category | | | | Υ | | |
| All ECG Values for Subjects with a Value of PCI | | | Υ | | | |
| ECG Values of PCI | | | Υ | | | |
| Abnormal ECG Findings | | | Υ | | | |
| Vital Signs | | | | | | |
| Vital Signs by Visit | Υ | | | Υ | | |
| Emergent Vital Signs Results by PCI Criteria | Υ | | | | | |
| All Vital Signs for Subjects with Values of PCI | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8. SECONDARY STATISTICAL ANALYSES

#### 8.1. Plasma Pharmacokinetic Analyses

## 8.1.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic" population, unless otherwise specified. There are no planned statistical analyses.

GUI\_51487 (4.0), effective October 2014, contains the pharmacokinetic methods to be used in non-compartmental analysis (NCA) and reporting of pharmacokinetic studies. This document should be used as a reference.

#### 8.1.2. Overview of Planned pharmacokinetic Analyses

Table provides an overview of the planned pharmacokinetic analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 8 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Untrans | formed | | | Log-transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Summai | γ | Individua | al | Summa | 'n | Individu | al |
| | Т | F | F | L | Т | F | F | L |
| Pharmacokinetic | | | | | | | | |
| Plasma Drug concentration | Υ | <b>Y</b> [1][2] | <b>Y</b> [1] | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = represents FL related to any displays of individual subject observed raw data.
- [1]: Linear and Semi-Log plots will be created on the same display.
- [2]: Separate Mean (± SD) and Median plots will be generated.

#### 8.1.3. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions, Section 11.4.3 Reporting process & standards for details on how the concentration data will be derived.

#### 8.1.3.1. Statistical Analysis of Pharmacokinetic Parameters

No formal pharmacokinetic statistical analyses will be performed.

#### 8.2. Pharmacodynamic/Biomarker Analyses

The pharmacodynamic/biomarker analyses will be based on the "Safety" population, unless otherwise specified.

#### 8.2.1. Overview of Planned Analyses

Table 10 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 10 Overview of Planned Pharmacodynamic/biomarker Analyses

| Endpoint | | | A | Absolu | ite | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Individual | | Stats Analysis | | | Summary | | Indiv | idual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Pharmacodynamic and Biomarkers | | | | | | | | | | | | | | |
| Inflammatory<br>biomarkers in skin<br>biopsy <sup>1</sup> | | | | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | | | |
| mRNA from skin biopsy <sup>2</sup> | | | | Υ | | Υ | Υ | Υ | Υ | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data
- 1: Histopathloogical Scoring of Skin biopsy may include epidermal thickness, elastase positive dermal cells, K16, CD3/CD11c and CD161.
- 2: mRNA expression of inflammatory gene transcripts including but not limited to:IL-4, IL-10, IL-17, IL-21, IL-22, IL-23, TNF, IFNy

# 8.2.2. Statistical Analysis of Inflammatory Biomarkers in the Skin Biopsy (Histopathological Scoring of Psoriatic Lesional Biopsies)

## Primary Statistical Analyses

#### Endpoint(s)

• Change from baseline on log transformed inflammatory biomarkers from skin biopsy on Day 43 pre-dose: Loge Change = Loge (Visit) – loge (Baseline)

#### Model Specification

- Endpoints will be statistically analyzed using an Analysis of Covariance (ANCOVA) model.
- Terms fitted in the ANCOVA model will include:
  - Fixed Category : Treatment
  - o Fixed Continuous Covariates : Loge Baseline score

#### **Model Checking & Diagnostics**

Refer to Appendix 1: Model Checking and Diagnostics for Statistical Analyses.

#### Presentation of results

#### **Primary Statistical Analyses**

- Adjusted geometric means, the mean difference between each dose (test) and the placebo (reference) at each timepoint and associated 95% confidence interval will be constructed using the residual variance
- ➤ The treatment ratios and 95% CI will be calculated by back-transforming the difference between the least square means and associated 95% CI
- ➤ Percentage change from baseline at each timepoint will be calculated from the adjusted geometric means using the formula 100% x (exp(adj mean)- 1)

## 8.2.3. Statistical Analysis of mRNA from Skin Biopsies: Transcriptomic Data

#### 8.2.3.1. Fold Change Analysis

The log<sub>2</sub> normalised copy numbers (also referred to as log2(intensity)) received from the normalised process will be listed and summarised appropriately.

As the data will be  $log_2$  transformed prior to the analysis the treatment effects will be expressed as ratios after back transformation to the original scale. These ratios can be converted from treatment ratios to fold change values as follows:

- If ratio  $\geq 0$  then fold change = ratio
- If ratio <0 then fold change = -1/ratio

#### **Primary Statistical Analyses**

#### Endpoint(s)

 Log2(intensity) mRNA expression of inflammatory gene transcripts which may include, but are not limited to the following as data permit: IL-4, IL-10, IL-17, IL-21, IL-22, IL-23, TNF and IFNy

#### **Model Specification**

- Endpoints will be statistically analyzed using a linear repeated measures mixed effects model.
- Terms fitted in the linear repeated measures mixed effects model will include:

Fixed Category : Treatment, Visit, Treatment \* Visit

Random Effect : Subject

#### **Model Checking & Diagnostics**

Refer to Appendix 1: Model Checking and Diagnostics for Statistical Analyses.

#### **Presentation of Results**

- For each probeset analysed adjusted means with corresponding 95% CI and fold changes with corresponding 95% CI's can be outputted. The fold change is derived from the ratio of the back-transformed estimate of the difference between adjusted means.
- Plots of LS means and 95% confidence intervals from the model will be generated for each treatment by time. Additionally, plots of differences and 95% confidence intervals for the comparison between the treatment groups will be generated.

For each comparison subsets of probesets will be identified based on an appropriate fold-change, for example, fold changes >1.5 or <-1.5. The proportion of probesets with fold changes >1.5 or <-1.5 will be summarised in a frequency table.

Exploratory graphical reporting on the back-transformed scale can include:

- Log<sub>2</sub> (intensity) plotted against time point separately for individual subjects, grouped by treatment group
- Adjusted mean intensity and 95 CI% plotted by treatment group and time point

## 8.3. Efficacy Analyses

#### 8.3.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the "Safety" population, unless otherwise specified.

Table 11 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 11 Overview of Planned Efficacy Analyses

| ENDPOINT | | | Α | bsolu | te | | % Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | | Sumi | mary | Individual | | Stats Analysis | | | Sumi | mary | Individual | |
| | T | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Psoriatic Lesion Severity Sum (PLSS) | | | | | | | | | | | | | | |
| PLSS | | | | Υ | Υ | Υ | Υ | Y | Y | Υ | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.3.2. Statistical Analysis of Efficacy Data

#### Statistical Analyses

#### Secondary Endpoint(s)

Percentage change from baseline (pre-dose Day 1) in PLSS score at Days 15, 29, 43 (pre-dose), 57, 71 and 85.

#### **Model Specification**

- Endpoints will be statistically analyzed using a mixed models repeated measures (MMRM) approach.
- Terms fitted in the MMRM model will include:
  - Fixed Category : Treatment, Day, Treatment\*Day

Clinical Study Identifier

#### **Statistical Analyses**

o Fixed Continuous Covariates : Baseline Score

Repeated Effect : Day

Note: Other covariates maybe explored, if deemed appropriate for sensitivity analyses.

#### **Model Checking & Diagnostics**

• Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### Presentation of results

- LS means and corresponding standard error of means (SEs) and 95% confidence intervals will be presented for each treatment by time interaction, together with estimated treatment differences (GSK2982772 – Placebo) and the corresponding 95% confidence intervals will be produced.
- Plots of LS means and 95% confidence intervals from the model will be generated over time by treatment. Additionally, plots of differences and 95% confidence intervals for the comparison of interest will be generated over time.

#### 9. OTHER STATISTICAL ANALYSES

#### 9.1. Skin Pharmacokinetic Analyses

#### 9.1.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic" population, unless otherwise specified. There are no planned statistical analyses.

GUI\_51487 (4.0), effective October 2014, contains the pharmacokinetic methods to be used in non-compartmental analysis (NCA) and reporting of pharmacokinetic studies. This document should be used as a reference.

## 9.1.2. Overview of Planned pharmacokinetic Analyses

Table provides an overview of the planned pharmacokinetic analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 8 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Untrans | formed | | | Log-transformed | | | |
|---|---|---|---|---|---|---|---|---|
| | Summai | Ύ | Individua | al | Summa | 'n | Individu | al |
| | Т | F | F | L | Т | F | F | L |
| Pharmacokinetic | | | | | | | | |
| Skin Drug concentration | Υ | <b>Y</b> [1][2] | <b>Y</b> [1] | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = represents FL related to any displays of individual subject observed raw data.
- [1]: Linear and Semi-Log plots will be created on the same display.
- [2]: Separate Mean (± SD) and Median plots will be generated.

#### 9.1.3. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions, Section 11.4.3 Reporting process & standards for details on how the concentration data will be derived.

#### 9.1.3.1. Statistical Analysis of Pharmacokinetic Parameters

No formal pharmacokinetic statistical analyses will be performed.

## 9.2. Exploratory Pharmacodynamic and Biomarker Analyses

The Biomarker analyses will be based on the "Safety" population, unless otherwise specified.

Clinical Study Identifier

Table 13 provides an overview of the planned Pharmacodynamic/Biomarker analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

Table 13 Overview of Planned Exploratory Biomarker Analyses

| Endpoint | | | ļ | Absolu | ite | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Τ | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Pharmacodynamic and Biomarkers | | | | | | | | | | | | | | |
| Inflammatory<br>biomarkers in blood <sup>1</sup> | | | | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | | | Υ |
| Target Engagament<br>Assay RIP1 (TEAR1) <sup>2</sup> | Υ | Υ | Υ | Υ | | Υ | Υ | | | | | | | |
| Pharmacology biomarker in skin <sup>3</sup> | | | | | | | | | | | | | | |
| Blood Transcptomics sample 4 | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1: Including, but not limited to CRP, VEGF, S100A8, IL-17, IL-22 and TNF
- 2: In blood and skin
- 3: Total or phosprylated RIP1, MLKL, and RIP3, cleaved and total caspase 8 signatures are not intended to be delivered as part of DBF by first intent. Any future summaries and/or analyses will be deemed post-hoc
- 4. Transcriptomic analysis of mRNA are not intended to be delivered as part of DBF by first intent. Any future summaries and/or analyses will be deemed post-hoc.

Scatter plots of Skin Target Engagement and skin biomarkers for Day 43 and Day 85 will also be produced.

If deemed appropriate, the relationship between Skin Target Engagement and the skin biomarkers will be explored further using multivariate statistical analyses. The consistency in the changes over time between the endpoints will also be assessed. Any such analyses will be defined after unblinding of the data and thus deemed post-hoc.

## 9.2.1. Planned Exploratory Biomarker Statistical Analyses

## Planned Statistical Analyses

#### Endpoint(s)

 Percentage change from baseline in blood inflammatory markers, including, but not limited to the following as data permits: CRP, VEGF, S100A8, IL-17, IL-22 and TNF across Days 43 (pre-dose) and 84 (pre-dose).

#### **Model Specification**

 Change from baseline scores will be analysed using a mixed models repeated measures (MMRM) across Day 43(pre-dose) and 85.

Clinical Study Identifier

#### **Planned Statistical Analyses**

Terms fitted in the MMRM model will include:

Fixed Category : Treatment, Day, Treatment\*Day

Fixed Continuous effect : Baseline scores

Repeated Effect : Day

#### **Model Checking**

• Refer to Appendix 1: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted means and corresponding standard error of means (SEs) and 95% confidence intervals will be presented for each treatment by time interaction, together with estimated treatment differences (GSK2982772 – Placebo) and the corresponding 95% confidence intervals will be produced for respective endpoints.
- Plots of LS means and 95% confidence intervals from the model will be generated for each treatment by time. Additionally, plots of differences and 95% confidence intervals for the comparison of interest will be generated.

#### **Target Engagement**

#### **Endpoints**

• Log Ratio = Log (free TEAR1) – log (total TEAR1)

#### **Model Specification**

- A mixed effect model will be fitted with treatment, period, time (i.e. planned relative time) and treatment \* time as a fixed effect and subject as a random effect. Baseline log ratio will be fitted as a continuous covariate
- The Kenward & Roger (KR) degrees of freedom approach will be used.

#### **Model Checking**

Refer to Section 11.11.

#### **Presentation of Results**

- Adjusted geometric means, the mean difference between each dose (test) and the placebo (reference) at each timepoint and associated 95% confidence interval will be constructed using the residual variance
- ➤ The treatment ratios and 95% CI will be calculated by back-transforming the difference between the least square means and associated 95% CI
- ➤ Percentage target engagement at each timepoint will be calculated from the adjusted geometric means using the formula 100% x (exp In (v2 / v1) 1) percentage target engagement = (100 engagement ratio) \* 100

## 9.3. Exploratory Efficacy Analyses

The exploratory efficacy analyses will be based on the "Safety" population, unless otherwise specified.

Table 14 provides an overview of the planned exploratory efficacy analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 14 Overview of Planned Exploratory Efficacy Analyses

| Endpoint(s) | | | Α | bsolu | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Anal | ysis | Sum | mary | Indiv | idual | Sta | ts Ana | lysis | Summary | | Indiv | ridual |
| | Т | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| Psoriasis Area Severity Index (PASI) | | | | | | | | | | | | | | |
| PASI score | | | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | Υ |
| PASI50, PASI75, | Υ | | Υ | Υ | | | Υ | | | | | | | |
| PASI90 <sup>1</sup> | | | | | | | | | | | | | | |
| Physician Global Asses | ssmei | nt (PG | A) | | | | | | | | | | | |
| PGA | | | | Υ | Υ | | Υ | Υ | | Υ | Υ | | | Υ |
| PGA (clear vs almost | Υ | | Υ | Υ | | | Υ | | | | | | | |
| clear) | | | | | | | | | | | | | | |
| Psoriatic Body Surface | Area | | | | | | | | | | | | | |
| BSA | | | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | Υ |
| Patient Reported Outco | omes | (PROs | 5) | | | | | | | | | | | |
| Dermatology Life | | | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | Υ |
| Quality Index (DLQI) | | | | | | | | | | | | | | |
| Visual Analogue Scale | | | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | | Υ |
| (VAS) itch score | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- PASI 50/75/90 will only be analysed if >50% of subjects have a BSA >5% at baseline

#### 9.3.1. Planned Exploratory Efficacy Statistical Analyses

GEE modelling will only be performed if at least 30% response rate and Day 43 or Day 85 for any one treatment group. Further the proportion of subjects achieving PASI50/75/90 will only be performed if >50% of subjects have a BSA >5% at baseline.

#### **Exploratory Endpoint(s)**

- Proportion of subjects who achieve ≥ xx% improvement from baseline in PASI score at Days 15, 29, 43 (pre-dose), 57, 71 and 85 (if sufficient number of subjects are enrolled with a >5% BSA).
- Proportion of subjects who have a PGA score of 'clear' (0) or 'almost clear' (1) at Days 15,29,

Clinical Study Identifier

43(pre-dose), 57, 71 and 85.

#### **Model Specification**

- Will be analysed using a GEE (Generalized Estimating Equations) model across Day 15, 29, 43 (pre-dose), 57, 71 and 85.
- Terms fitted in the GEE model will include:

Fixed Category : Treatment, Day, Treatment\*Day

Repeated Effect : Day

#### Presentation of results

- Adjusted Odds Ratios and corresponding 95% confidence intervals will be generated from contrasts for treatment by day interactions.
- Plots of the adjusted Odds Ratios and 95% confidence intervals from the model will be generated for each treatment by time. Additionally plots of differences and 95% confidence intervals for the comparisons of interest will be generated.

#### **Exploratory Endpoint(s)**

- Psoriasis Area Severity Index (PASI) score (if sufficient number of subjects are enrolled with a >5% BSA).
- Physician Global Assessment (PGA)
- Visual Analogue Scale (VAS) itch score.

#### **Model Specification**

- Change from baseline scores will be analysed using a mixed models repeated measures (MMRM) across Day 15, 29, 43 (pre-dose), 57, 71 and 85.
- Terms fitted in the MMRM model will include:

Fixed Category : Treatment, Day, Treatment\*Day

Fixed Continuous effect : Baseline scores

Repeated Effect : Day

Note: Other covariates maybe explored, if deemed appropriate for sensitivity analyses.

#### **Presentation of results**

- Adjusted means and corresponding standard error of means (SEs) and 95% confidence intervals will be presented for each treatment by time interaction, together with estimated treatment differences (GSK2982772 – Placebo) and the corresponding 95% confidence intervals will be produced for respective endpoints.
- Plots of LS means and 95% confidence intervals from the model will be generated for each treatment by time. Additionally, plots of differences and 95% confidence intervals for the comparison of interest will be generated.

#### **Exploratory Endpoint(s)**

Body Surface Area (BSA)

#### Model Specification

- Change from baseline scores will be analysed using an Analysis of Covariance (ANCOVA) model at Day 85.
- Terms fitted in the ANCOVA model will include:

Fixed Category : TreatmentFixed Continuous effect : Baseline scores

#### Presentation of results

- Adjusted means and corresponding standard error of means (SEs) and 95% confidence intervals will be presented for each treatment, together with estimated treatment differences (GSK2982772 – Placebo) and the corresponding 95% confidence intervals will be produced.
- Plots of LS means and 95% confidence intervals from the model will be generated for each treatment. Additionally, plots of differences and 95% confidence intervals for the comparison of interest will be generated.

#### **Exploratory Endpoint(s)**

Dermatology Life Quality Index (DLQI) score.

#### **Model Specification**

- Change from baseline scores will be analysed using a mixed models repeated measures (MMRM) across Day 43 (pre-dose) and 85.
- Terms fitted in the MMRM model will include:

Fixed Category : Treatment, Day, Treatment\*Day

Fixed Continuous effect : Baseline scores

Repeated Effect : Day

#### Presentation of results

- Adjusted means and corresponding standard error of means (SEs) and 95% confidence intervals will be presented for each treatment by time interaction, together with estimated treatment differences (GSK2982772 – Placebo) and the corresponding 95% confidence intervals will be produced for respective endpoints.
- Plots of LS means and 95% confidence intervals from the model will be generated for each treatment by time. Additionally, plots of differences and 95% confidence intervals for the comparison of interest will be generated.

#### **Model Checking**

Refer to Appendix 1: Model Checking and Diagnostics for Statistical Analyses.

## 9.4. Exploratory Pharmacodynamic / Efficacy Analyses

If deemed appropriate, the relationship between the skin biomarkers and efficacy endpoints will be explored further using multivariate statistical methods and/or Bayesian methodology as recommended by the GSK PCPS Experimental Medicine working group. The consistency in the changes over time between the endpoints will also be assessed. Any such analyses will be defined after unblinding of the interim data and thus deemed post-hoc.

## 10. REFERENCES

## 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.1 | Appendix 1: Time and Events |
| Section 11.2 | Appendix 2: Assessment Windows |
| Section 11.3 | Appendix 3: Treatment States & Phases |
| Section 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| Section 11.5 | Appendix 5: Derived and Transformed Data |
| Section 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| Section 11.7 | Appendix 7: Values of Potential Clinical Importance |
| Section 11.8 | Appendix 8: Multicentre Studies |
| Section 11.9 | Appendix 9: Examination of Covariates and Subgroups |
| Section 11.10 | Appendix 10: Multiple Comparisons and Multiplicity |
| Section 11.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP Appendices | |
| Section 11.12 | Appendix 12: Abbreviations & Trade Marks |
| Section 11.13 | Appendix 13: List of Data Displays |
| Section 11.14 | Appendix 14: Example Mock Shells for Data Displays |

## 11.1. Appendix 1: Time & Events

## 11.1.1. Protocol Defined Time & Events

| | | Treatment Period | | | | | | | Notes | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening | | | | | | | | | | | | | Day 85 | Ear | | $85 \pm 2$ d. Early Withdrawal: NA Follow Up: 28d after last dose $\pm$ 3d |
| Screening<br>Procedures | exclu | Screening procedures in addition to those listed below are (outpatient visit): informed consent; inclusion/exclusion criteria; demography; medical history (includes past and current conditions, medication history, a amily history of premature CV disease); HIV, Hep B and Hep C screen; serum pregnancy test (WCBP only | | | | | | | | | s, medication history, and | | | | | | |
| Site Visit | Х | X | X | Х | lataro | X | loode | X | , , , | X | 11011 | X | 00.00 | X | Х | Х | 1. Full physical exam: |
| Phone call | | | | | Х | | Х | | Χ | | Х | | Х | | | | height/weight at |
| Safety Assessme | ents | | | | | | | | | | | | | | | | Screening, height not<br>required at later |
| Full physical exam <sup>1</sup> | Х | | | | | | | | | | | | | Х | Х | Х | timepoints. 2. Vitals: BP, HR, RR, |
| Brief physical exam | | X<br>5 | | Х | | Х | | X<br>5 | | Х | | Х | | | | | temperature. ECG<br>triplicate at Screening<br>only. |
| 12-lead ECG,<br>vital signs² | Χ | <b>X</b> 5 | Х | Х | | Χ | | X<br>5 | | Х | | Х | | Х | Х | Х | 3. Urinalysis not required on Days 29, 57 and 71. |
| Columbia Suicide<br>Severity Rating<br>Scale (C-SSRS) | х | <b>X</b> 5 | | | | | | X<br>5 | | | | | | х | х | | 4. If urine test is positive, confirmatory serum test must be performed. |
| Hematology,<br>chemistry,<br>urinalysis | Х | X<br>5 | Х | Х | | X<br>3 | | X<br>5 | | X<br>3 | | X3 | | Х | Х | Х | 5. Pre-dose 6. In Cohort 1, subjects must take study medication twice a day |
| FSH & estradiol (if applicable) | Х | | | | | | | | | | | | | | | | approx. 12h apart. In Cohort 2, subjects must |
| Serum<br>pregnancy<br>(WCBP) | Х | | | | | | | | | | | | | | | | take study medication<br>three times a day<br>approx. 8h apart. Exact<br>time of dosing to be |
| Urine pregnancy<br>test (WCBP<br>only) <sup>4</sup> | | X<br>5 | Х | Х | | Х | | X<br>5 | | Х | | Х | | Х | Х | Х | subjects must not take |
| Study Treatment | | | | | | | | | medication at home in<br>the morning. Subjects | | | | | | | | |
| Randomisation | | Х | | | | | | | | | | | | | | | will complete pre-dose<br>assessments and then<br>will be administered their |
| Study<br>medication <sup>6</sup> | | Х | X | | | | | | | X | , | | | | - | | |
| Dispensing of study medication | | Х | | | | Χ | | | | Χ | | | | | | | morning dose of<br>medication at site on<br>Day 43 only. On Day 85, |
| Dispensing of diary cards <sup>7</sup> | | Х | Χ | Χ | | Χ | | Х | | Х | | Х | | | | | subjects no longer dosed. |

Clinical Study Identifier **Treatment Period Notes** Visit windows Screening: up to 30d Early Withdrawal 14 before Day 1. Treatment Period Day 43 Day 50 Day 15 Day 29 Day 85 **Day 22** Day 36 Day 57 Day 64 Day 71 Day /8 **Procedures** Day 8 Day 1 (except Day 1 & 85):  $\pm$  3d. Day 1 NA; Day  $85 \pm 2d$ . Early Withdrawal: NA Follow Up: 28d after last dose  $\pm$  3d 7. Diary card checked by PROs/ Disease Assessments site staff and new diary Psoriatic Body Χ Χ Χ Χ card dispensed at every 5 Surface Area study visit. PASI, PGA. Χ Χ Χ Χ 8. Blood samples for Χ Χ Χ Χ Χ 5 PLSS, Itch inflammatory biomarkers and mRNA taken pre-Χ Χ Χ Χ Χ DLQI dose on Day 1, Day 43 5 5 and Day 85. Photograph of Χ Χ Χ Χ 9. PK blood samples lesions 5 taken pre-dose on Day 43. Post-dose serial PK Other Assessments and Procedures samples taken on Day 1 Blood sample for Χ Χ and Day 43 at 1, 2, 4, Χ Χ inflammatory 5 5 and 6 hours post-dose. biomarkers8 10. Pre-dose Day 1 one Blood sample for Χ Χ biopsy taken from non-Χ Χ 5 mRNA analysis8 lesional skin and two biopsies taken from Blood sample for Χ Χ biopsy target lesion. Χ Χ Target 5 5 11. On Day 43, two Engagement biopsies taken from the PK blood Χ Χ Χ same target lesion that Χ samples9 5 was selected at Day 1. Skin punch Punch biopsies on Day 43 are to be taken prebiopsies for PK, dose. inflammatory Χ 12. Biopsy only required biomarkers, Χ 5,1 X12 at Early Withdrawal visit 11 mRNA, target 0 if completed at least 14 engagement & days of treatment and pathway prior to Day 43. engagement 13. PGx sample Pharmacogenetic Χ collected at Day 1. after sample (PGx) randomization and separate informed consent. If sample not collected at Day 1, can be collected at any time post-randomization. Con med review 14. If subject withdraws & AE/SAE early, every effort will be reporting made for the subject to complete an Early Withdrawal visit prior to Follow Up.

## 11.2. Appendix 2: Assessment Windows

## 11.2.1. Definitions of Assessment Windows for Analyses

No Assessment Windows will be defined for Analysis, and summaries and analyses will be based on nominal visits.

## 11.3. Appendix 3: Treatment States and Phases

#### 11.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment unless otherwise specified. Treatment phases are to be included on A&R datasets.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date |
| Post-Treatment | Date > Study Treatment Stop Date |

#### 11.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 11.3.2.1. Treatment States for Safety Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date +1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### **Treatment States for AE Data**

| Treatment State | Definition |
|---|---|
| AE = Pre-Treatment | AE Start Date < Study Treatment Start Date |
| AE = On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date +1 |
| AE = Post-Treatment | If AE onset date is after the treatment stop date. AE Start Date > Study Treatment Stop Date |
| AE Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date: <b>= AE Onset Date - Treatment Start Date</b> If Treatment Start Date ≤ AE Onset Date: <b>= AE Onset Date - Treatment Start Date +1</b> Missing otherwise. |
| AE Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| AE = Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing]. |

#### NOTES:

If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 11.4. Appendix 4: Data Display Standards & Handling Conventions

#### 11.4.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order [1] |
| Α | GSK2982772 60mg BID | GSK2982772 60mg BID | 2 |
| С | GSK2982772 60mg TID | GSK2982772 60mg TID | 3 |
| Р | Placebo | Placebo [2] | |
| Q | Placebo TID | Flacebo (4) | |

#### NOTES:

- 1. Order represents treatments being presented in TFL, as appropriate.
- 2. Placebo BID and Placebo TID will be combined for reporting purposes

Should a subject receive the wrong medication at any point during the study in error, that subject will be treated as having received GSK2982772 60mg BID or GSK2982772 60mg TID, dependent on whether Cohort 1 or Cohort 2, for the duration of the study. Such subjects will have a footnote on Table 1.12 and Listing 1.

#### 11.4.2. Baseline Definition & Derivations

#### 11.4.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

| Parameter | Study Assessmen | Baseline Used in | | | | | | | |
|---|---|---|---|--|--|--|--|--|--|
| | Screening | Day 1 (Pre-Dose) | Data Display | | | | | | |
| Safety Assessments | Safety Assessments | | | | | | | | |
| Vital signs <sup>1</sup> | X | X | Day 1 (Pre-Dose) | | | | | | |
| 12-lead ECG <sup>2</sup> | X | X | Day 1 (Pre-Dose) | | | | | | |
| Laboratory<br>(Haematology,<br>clinical chemistry and<br>urinalysis) | X | X | Day 1 (Pre-Dose) | | | | | | |
| Columbia Suicide<br>Severity Rating<br>Scale (C-SSRS) | X | X | Day 1 (Pre-Dose) | | | | | | |
| PROs/Disease Assessments | | | | | | | | | |
| Psoriatic Body | X | X | Day 1 (Pre-Dose) | | | | | | |
| Parameter | Study Assessments Considered As Baseline | | Baseline Used in |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | Data Display |
| Surface Area | | | |
| PASI, PGA, PLSS, itch | X | X | Day 1 (Pre-Dose) |
| DLQI | Х | X | Day 1 (Pre-Dose) |
| Other Assessments a | and Procedures | | |
| Blood sample for inflammatory biomarkers | | X | Day 1 (Pre-Dose) |
| Blood sample for mRNA analysis | | X | Day 1 (Pre-Dose) |
| Blood sample for<br>Target Engagement | | X | Day 1 (Pre-Dose) |
| PK blood samples | | Х | Day 1 (Pre-Dose) |
| Skin punch biopsies<br>for PK, inflammatory<br>biomarkers, mRNA,<br>target engagement &<br>pathway<br>engagement | | X | Day 1 (Pre-Dose) |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- 1 = Vitals: BP, HR, RR, temperature
- 2 = ECG triplicate at screening only

#### 11.4.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from | = Calculate the change from baseline at each given timepoint |
| Baseline | and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.4.2.1 Baseline Definitions will be
  used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 11.4.3. Reporting Process & Standards

| Reporting Process |
|-------------------|
| Software |

| Reporting Process | |
|---|---|
| The currently support the currently support to the currently suppo | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | UK1SALX00175 |
| HARP Area | arenv \ arprod \ gsk2982772 \ mid203167 \ internal_03 |
| | arenv \ arprod \ gsk2982772 \ mid203167 \ final |
| QC Spreadsheet | arenv \ arprod \ gsk2982772 \ mid203167 \ internal_03 |
| | arenv \ arwork \ gsk2982772 \ mid203167 \ final \ documents |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to Integrated Data Standards Library (IDSL)<br/>GSK A&amp;R dataset standards.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for key outputs at the time of the IA, SAC. | |

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

| Reporting Standard | Reporting Standards |
|---|---|
| • Unscheduled visits will not be included in summary tables or figures, unless otherwise stated | |
| All unscheduled v | All unscheduled visits will be listed. |
| <b>Descriptive Summa</b> | ry Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharm | acokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and [between and or within] geometric coefficient of variation (CVb/w (%)) will be reported.</li> <li>[1] CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data)</li> <li>[2] CV<sub>w</sub> (%) = √ (exp(MSE) - 1) * 100 (MSE = mean square error from mixed effect model of loge-transformed data).</li> </ul> |
| Parameters Not<br>Being Log<br>Transformed | tmax, first point, last point and number of points used in the determination of Lambda_z. |
| Summary Tables | The following PK parameters will not be summarised: tmax, first point, last point and number of points used in the determination of Lambda_z. |
| Listings | Additionally, include the first point, last point and number of points used in the determination of lambda_z for listings. |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing 
    → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### 11.5.2. Study Population

#### **Demographics**

#### Date of Birth

Only the year of birth will be captured, and therefore the date of birth is then derived as follows:
 Year of birth = YYYY → Date of birth = 30th June YYYY

#### Age

- Calculated as the integer part of (date of baseline date of birth)
   Age = integer part (date of baseline 30<sup>th</sup> June YYYY)
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>

#### Race category

- White: 'White: Arabic/North African Heritage' and 'White: White/Caucasian/European Heritage', or both of these, but no other category checked
- African descent: 'African American/African Heritage', and no other category checked
- Asian: 'Asian Central/South Asian Heritage', 'Asian East Asian Heritage', 'Asian Japanese Heritage', and 'Asian – South East Asian Heritage', or any combination of these, but no other category checked
- Other: Any combination that has not been categorized above ('mixed race')

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### **Extent of Exposure**

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

## 11.5.3. Safety

#### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

# **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - $\circ$  Example 3: 0 Significant Digits = '< x' becomes x 1

#### 11.5.4. Pharmacokinetic

#### **Skin Pharmacokinetic Concentrations**

#### Skin PK Conc

- The density of human skin tissue is 1.184 g/mL per Gastroplus V9.0.
- The volume of solvent added to each tissue sample was 0.5 mL.
- For actual tissue weights, please refer to the Excel spreadsheet

Skin PK Concentration (ng/mL)

- 1. PK Conc in Weight of Tissue Sample = SMS PK Conc in Soln (ng/mL) X [0.5 mL + (Tissue Weight (g) / 1.184 g/mL)]
- 2. PK Conc in tissue as concentration (ng/g) = PK Conc in Weight of Tissue Sample / Tissue Weight
- 3. PK Conc in tissue as concentration (ng/mL) = PK Conc in tissue as concentration (ng/g) 1.184 g/mL

Example (fictitious) data:

SMS tissue homogenate concentration = 2 ng/mL

Tissue weight = 0.014 g

SMS plasma concentration= 400 ng/mL

**Example Calculations:** 

- 1. Convert GSK2982772 concentration in the homogenate to GSK2982772 concentration in the tissue sample as follows:
- 2 ng/mL X  $[0.5 \text{ mL} + (0.014 \text{ g}/1.184 \text{ g/mL})] = 2 \text{ng/mL} \times 0.512 \text{ mL} = 1.024 \text{ ng GSK2982772}$  in a 0.014 g tissue sample
- 2. Convert absolute amount of GSK2982772 in this skin tissue sample to a tissue concentration as follows:
- 1.024 ng / 0.014 g tissue = 73.1 ng GSK2982772/g tissue = 73.1 ng/g
- Convert ng/g tissue to ng/mL tissue as follows :
- 73.1 ng/g X 1.184 g/mL = 86.5 ng GSK2982772/mL tissue = 86.5 ng/mL
- 4. Determine the ratio of GSK2982772 tissue concentration to GSK2982772 plasma concentration for a given patient as follows:
- 86.5 ng/mL / 400 ng/mL = 0.216

#### 11.5.5. Efficacy

#### **Clinical Efficacy**

# Plaque Lesional Severity Score (PLSS) and index plaque selection

Two plaques will be selected at Day -1, one for clinical assessment (index plaque) and one for biopsy. Ideally the index plaque should be the most severe plaque. At a minimum each plaque will have an induration score of  $\geq 2$  (moderate or above) and a score of  $\geq 1$  in erythema and scaling, as detailed in the scoring list below. Each lesion must have a PLSS score of  $\geq 5$ . The PLSS is the sum of the erythema, scaling and induration. The PLSS assessment will be performed by the same qualified dermatologist throughout, wherever possible and will be scored using the same scale (0-4 point rating scale) as the PASI.

#### **Clinical Efficacy**

#### Psoriasis Area Severity Index (PASI), PASI50, PASI75, PASI90

Psoriatic lesions will be assessed using the PASI. The PASI assessment will be performed by the investigator or a suitably trained delegate, and whenever possible, the PASI assessments for an individual subject will be completed by the same assessor at all time-points. Each area of the body (head, upper extremities, trunk, lower extremities) will be assessed for the following symptoms: erythema, induration, scaling. A 0–4 point rating scale will be used, as follows:

- 0 = No symptom
- 1 = Slight
- 2 = Moderate
- 3 = Marked
- 4 = Very Marked

After calculating the BSA as detailed above, use the multiplier for that body region to calculate the area score for each region as detailed below:

Head

Number of palms x 10% = % of head

Upper extremities

Number of palms x 5% = % of upper extremities

• Trunk

Number of palms x 3.3% = % of area trunk

Lower extremities

Number of palms x 2.5% = % of lower extremities

The area of psoriatic involvement for each area of the body (head, upper extremities, trunk, lower extremities) will be assessed using a 0–6 point rating scale, as follows:

- 0 = 0%
- 1 = 0 9%
- 2 = 10 29%
- 3 = 30 49%
- 4 = 50-69%
- 5 = 70-89%
- 6 = 90 100%

Total PASI score will be calculated using the following method:

- Add up the 3 intensity scores for each area of the body to give 4 subtotals (A1—A4):
  - A1 (head intensity score) = head redness score + head thickness score + head scaling score

#### **Clinical Efficacy**

- **A2** (upper extremities intensity score) = upper extremities **redness** score + upper extremities **thickness** score + upper extremities **scaling** score
- A3 (trunk intensity score) = trunk redness score + trunk thickness score + trunk scaling score
- A4 (lower extremities intensity score) = lower extremities redness score + lower extremities thickness score + lower extremities scaling score
- Multiply each subtotal (A1–A4) by the body surface area represented by that region to give 4 new subtotals (B1–B4):

B1 (head) = A1 x 0.1
 B2 (upper extremities) = A2 x 0.2
 B3 (trunk) = A3 x 0.3
 B4 (lower extremities) = A4 x 0.4

• Multiply each subtotal (B1–B4) by the area affected for that region to give 4 new subtotals (C1–C4):

C1 (head) = B1 x 1-6
 C2 (upper extremities) = B2 x 1-6
 C3 (trunk) = B3 x 1-6
 C4 (lower extremities) = B4 x 1-6

Calculate the total PASI score = C1 + C2 + C3 + C4

From the total scores, the following will be derived: change from baseline, percentage change from baseline, PASI50, PASI75 and PASI90 at each time point. Calculation of change from baseline and percentage change from baseline is described in Section 11.4.2.2.

Where PASI50, PASI75 and PASI90 are given by:

| PASI50 | Yes: | ≥ 50% reduction in PASI total score from baseline at time point |
|---|---|---|
| | No: | < 50% reduction in PASI total score from baseline at time point |
| PASI75 | Yes: | ≥ 75% reduction in PASI total score from baseline at time point |
| | No: | < 75% reduction in PASI total score from baseline at time point |
| PASI90 | Yes: | ≥ 90% reduction in PASI total score from baseline at time point |
| | No: | < 90% reduction in PASI total score from baseline at time point |

#### Physician Global Assessment (PGA)

Psoriatic lesions will be assessed using the PGA. The PGA assessment will be performed by the investigator or a suitably trained delegate, and whenever possible, the PGA assessments for an individual subject will be completed by the same assessor at all time-points. A 6-point scoring system will be used to measure the severity of psoriatic lesions over the whole body, at the time of the evaluation:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.



| PGA (clear and almost clear) | | |
|---|---|---|
| PGA is given | ven by: | |
| PGA | Clear (0):<br>Almost<br>Clear (1): | No signs of psoriasis (post-inflammatory hypopigmentation or hyperpigmentaition could be present) slight elevation, scale and/or erythema |

## **Body Surface Area (BSA)**

As part of the inclusion criteria the patients Psoarisis plaques need to cover 2-10% of body surface area. This will be calculated based on the areas outlined as part of the PASI score (see section 9.6.4.2). Where body surface area is calculated based on the palm method, where a patient's palm to PIP and thumb = 1%, and so:

| Head and Neck | 10% (10 palms) |
|------------------------------|----------------|
| Upper extremities | 20% (20 palms) |
| Trunk (axillae and groin) | 30% (30 palms) |
| Lower extremities (buttocks) | 40% (40 palms) |

Therefore the total BSA = 100% (100 palms)

So these proportions are applied to the absolute areas identified at Baseline to determine the overall body surface area, assuming that the areas are available. If only the categories are available (eg. 0-9%, 10-29%) then this calculation cannot be calculated.

#### **Dermatology Life Quality Index (DLQI)**

The Dermatology Life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above.

#### **CONFIDENTIAL**

Clinical Study Identifier

| Clinical Efficacy CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by |
|---|
| third party copyright laws and therefore have been excluded. |

### **Clinical Efficacy**

CCI

#### Visual Analogue Scale (VAS) itch score

The subject will be asked to rate the intensity of itch over the past week by marking a line on a 10 cm VAS with anchors "0" (no noticeable itching) to "10" (maximum itching sensation).

# 11.5.6. Pharmacodynamic and Biomarker

#### **TEAR**

## **Target Engagement**

- Ratio = free / total
- Target Engagement = 100 (ratio post/ratio baseline) \* 100))
- BIOMARK dataset: BICATCD = TRALBP1 (total) or RALB1F (free)

BITESTCD = CONC (Sample = Target Engagement) and CONCTSZ (Sample = Tru Culture)

# 11.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

## 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study at the discretion of the investigator.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and</li> </ul> |
| | figures, unless otherwise specified. |

# 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument : |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to</li> </ul> |
| | be missing data and should be displayed as such. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 11.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. Imputed dates should be stored in variables IMPSTDT (Imputed Start Date) and IMPENDT (Imputed End Date) |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |

# 11.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.6.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| PLSS | <ul> <li>Actual score: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time.</li> <li>Percentage change from baseline: <ul> <li>If baseline missing: Exclude from analysis</li> <li>If baseline not missing: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time</li> </ul> </li> </ul> |
| PASI | Change from baseline: If baseline missing: Exclude from analysis If baseline not missing: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time. |
| PASI50 | If the data is missing then failure is assumed, and therefore a 'non-response' |

| Element | Reporting Detail |
|---|---|
| PASI75<br>PASI90 | assigned to the missing data point. |
| PGA | <ul> <li>Actual score: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time.</li> <li>Change from baseline: <ul> <li>If baseline missing: Exclude from analysis</li> <li>If baseline not missing: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time.</li> </ul> </li> </ul> |
| PGA (clear and almost) | If the data is missing then failure is assumed, and therefore a 'non-response' assigned to the missing data point. |
| BSA | Change from baseline: If data is missing, exclude from analysis as it is not possible to calculate change from baseline since BSA is measured at only two time points; baseline (Day 1 pre-dose) and at Day 85. |
| DLQI | <ul> <li>Actual score: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time.</li> <li>Change from baseline: <ul> <li>If baseline missing: Exclude from analysis</li> <li>If baseline not missing: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time.</li> </ul> </li> </ul> |
| VAS | <ul> <li>Actual score: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time.</li> <li>Change from baseline: <ul> <li>If baseline missing: Exclude from analysis</li> </ul> </li> <li>If baseline not missing: The mixed models repeated measures model will be applied to the data in the analysis and account for missing data in the repeated measures analysis over time.</li> </ul> |

# 11.7. Appendix 7: Values of Potential Clinical Importance

# 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

#### 11.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| | | > 450 [1] | |
| Abaaluta OTa Intanial | | > 450 [2] | ≤ 479 <sup>[2]</sup> |
| Absolute QTc Interval | msec | ≥ 480 <sup>[2]</sup> | ≤ 499 <sup>[2]</sup> |
| | | ≥ 500 <sup>[2]</sup> | |
| Absolute PR Interval | msec | < 110 <sup>[1]</sup> | > 220 [1] |
| Absolute QRS Interval | msec | < 75 <sup>[1]</sup> | > 110 [1] |
| Change from Baseline | | | |
| | msec | > 60 [1] | |
| Increase from Baseline QTc | msec | > 30 [2] | ≤ <b>59</b> <sup>[2]</sup> |
| NATE OF THE PROPERTY OF THE PR | msec | ≥ 60 <sup>[2]</sup> | |

**NOTES:** [Remove footnotes for RAP development]

- 1. Represent standard ECG values of PCI for HV studies
- 2. Represent further subdivisions of ECG values for analysis whereby the RAP team needs to decide whether these need to be generated in addition to standard ECG values being flagged. IF not required, then delete.

### 11.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

**NOTES:** : [Remove footnotes for RAP development]

Represent further subdivisions of BP & HR for analysis whereby the RAP team needs to decide whether these need to be generated in addition to standard absolute BP & HR values being flagged. IF not required, then delete.

### CONFIDENTIAL

Clinical Study Identifier

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| 11.8. Appendix 8: Multicenter Studies | | | | | |

No specific outputs will be produced by centre or highlighting the recruitment by site.

# 11.9. Appendix 9: Examination of Covariates, Subgroups & Other Strata

No sub group analyses are to be conducted in this study.

# 11.10. Appendix 10: Multiple Comparisons & Multiplicity

No adjustments will be made for multiplicity.

# 11.11. Appendix 11: Model Checking and Diagnostics for Statistical Analyses

#### 11.11.1. Statistical Analysis Assumptions

## Analysis • MMRM

- For the MMRM, model assumptions will be applied, but appropriate adjustments maybe applied based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

# 11.12. Appendix 12 – Abbreviations & Trade Marks

# 11.12.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| IA, SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

# 11.12.2. Trademarks

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
| SAS |

# 11.13. Appendix 13: List of Data Displays

## 11.13.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacokinetic / Pharmacodynamic | 6.1 to 6.n | 6.1 to 6.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y t | 0 <b>Z</b> |

## 11.13.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix [X]: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 11.13.3. Deliverable [Priority]

| Delivery | Description |
|----------|------------------------------------------------|
| IA | Interim Analysis Statistical Analysis Complete |
| IA, SAC | Final Statistical Analysis Complete |

# 11.13.4. Study Population Tables

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition | ICH E3, GSK CTR, FDAAA, EudraCT | IA, SAC |
| 1.2. | All screened | ES6 | Summary of Reasons for Screen Failure | Journal Requirements | IA, SAC |
| 1.3. | Safety | NS1 | Summary of Number of Subjects by Centre | EudraCT | IA, SAC |
| Protoco | ol Deviation | | | | |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | IA, SAC |
| Popula | tion Analysed | | | | |
| 1.5. | Safety | SP1 | Summary of Study Populations and Exclusions | IDSL | IA, SAC |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, GSK CTR, FDAAA, EudraCT | IA, SAC |
| 1.7. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, GSK CTR, FDAAA,<br>EudraCT | IA, SAC |
| 1.8. | Safety | DM6 | Summary of Race and Racial Combination Details | ICH E3, FDA | IA, SAC |
| 1.9. | Safety | | Summary of Psoarsis Baseline Characteristics | Based on DM1 to include: Baseline BSA, Duration, Prior Treatment, Naive to Phototherapy, Baseline PASI Score, Baseline PLSS score, Baseline PGA, Lesion Seveirty (area and score), history of tobacco use | IA, SAC |
| Prior ar | nd Concomitan | t Medications | | | |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.10. | Safety | MH4 | Summary of Current/Past Medical Conditions | ICH E3 Separate summaries for Current & Past conditions, if collected. | IA, SAC |
| 1.11. | Safety | CM1 | Summary of Concomitant Medications | ICH E3 | IA, SAC |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.12. | Safety | EX1, EX2,<br>OEX1, OEX5 | Summary of Exposure to Study Treatment | ICH E3 Dose and/or time on treatment, as applicable. | IA, SAC |

# 11.13.5. Safety Tables

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | e Events (AEs) | | | | |
| 2.1. | Safety | AE5a | Summary of All Adverse Events by System Organ Class and Maximum Intensity | ICH E3 | IA, SAC |
| 2.2. | Safety | AE3 | Summary of Common (>10%) Adverse Events by Overall Frequency | GSK CTR | IA, SAC |
| 2.3. | Safety | AE5a | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Intensity | GSK CTR | IA, SAC |
| Serious | Serious and Other Significant Adverse Events | | | | |
| 2.4. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class | IDSL / GSK CTR | IA, SAC |
| 2.5. | Safety | CP_AE8a | Listing of Fatal Adverse Events | | IA, SAC |

| Safety : | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class | GSK CTR | IA, SAC |
| 2.7. | Safety | AE3 | Summary of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment by Overall Frequency | IDSL | IA, SAC |
| 2.8. | Safety | AE16 | Summary of Subjects and Number of Occurrences of Serious,<br>Drug-Related Serious, Fatal Serious, and Drug-Related Fatal<br>Serious Adverse Events | FDAAA, EudraCT | IA, SAC |
| Labora | tory: Chemistry | / | | | |
| 2.9. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline | ICH E3 Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | IA, SAC |
| 2.10. | Safety | LB1 | Summary of Clinical Chemistry Values | | IA, SAC |
| 2.11. | Safety | LB3 | Summary of Emergent Clinical Chemistry Results by Potential Clinical Importance Criteria | | IA, SAC |
| Labora | tory: Hematolo | gy | | | • |
| 2.12. | Safety | LB1 | Summary of Hematology Changes From Baseline | ICH E3 Includes baseline values. | IA, SAC |
| 2.13. | Safety | LB1 | Summary of Hematology Values | ICH E3 Includes baseline values. | IA, SAC |
| 2.14. | Safety | LB3 | Summary of Emergent Hematology Results by Potential Clinical Importance Criteria | | IA, SAC |
| Labora | tory: Urinalysis | <b>,</b> | | | |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.15. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3<br>Includes Baseline values. | IA, SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 2.16. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | IA, SAC |
| 2.17. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | IA, SAC |
| ECG | | | | | |
| 2.18. | Safety | EG1 | Summary of ECG Findings | IDSL As above for Chemistry, using ECG findings categories (and change from baseline categories, if applicable). | IA, SAC |
| 2.19. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | IA, SAC |
| 2.20. | Safety | CP_EG12 | Summary of Maximum Change from Baseline in QTc Values by Category | IDSL | IA, SAC |
| Vital Si | gns | | | | |
| 2.21. | Safety | VS1 | Summary of Change From Baseline in Vital Signs by Visit | ICH E3 Includes Baseline values. | IA, SAC |
| 2.22. | Safety | VS1 | Summary of Vital Signs by Visit | | IA, SAC |

# 11.13.6. Safety Figures

| Safety : | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events | | | | |
| 2.1. | Safety | AE10 | Plot of Common Adverse Events and Relative Risk | IDSL<br>Common defined as >10% | IA, SAC |
| Hepatol | Hepatobilary (Liver) | | | | |
| 2.2. | Safety | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT | | IA, SAC |
| 2.3. | Safety | LIVER9 | Scatter Ploy for Maximum ALT va Maximum Total Bilirubin | | IA, SAC |

# 11.13.7. Efficacy Tables

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PLSS | | | | | |
| 3.1. | Safety | EFF_T3 | Summary Statistics for PLSS scores by Treatment and Visit | | IA, SAC |
| 3.2. | Safety | EFF_T3 | Summary Statistics for % change from baseline PLSS scores by Treatment and Visit | | IA, SAC |
| 3.3. | Safety | EFF_T4 | Summary of Statistical Analysis Results for Percentage Change from Baseline PLSS score by Visit | | IA, SAC |
| PASI | | | | | |
| 3.4. | Safety | EFF_T3 | Summary Statistics for PASI scores by Treatment and Visit | | IA, SAC |
| 3.5. | Safety | EFF_T3 | Summary Statistics for Change from baseline PASI scores by Treatment and Visit | | IA, SAC |
| 3.6. | Safety | EFF_T4 | Summary of Statistical Analysis Results for Percentage Change from Baseline PASI score by Visit | | IA, SAC |
| 3.7. | Safety | EFF_T2 | Frequency: Proportion of subjects improving from baseline in PASI Score (PASI 50. PASI 75 and PASI 90) by Treatment and Visit | | IA, SAC |
| 3.8. | Safety | EFF_T1 | GEE adjusted odds ratio and 95% CI for PASI50 by Visit | | IA, SAC |
| 3.9. | Safety | EFF_T1 | GEE adjusted odds ratio and 95% CI for PASI75 by Visit | | IA, SAC |
| 3.10. | Safety | EFF_T1 | GEE adjusted odds ratio and 95% CI for PASI90 by Visit | | IA, SAC |
| PGA | | | | | |
| 3.11. | Safety | EFF_T3 | Summary Statistics for PGA Scores by Treatment and Visit | | IA, SAC |
| 3.12. | Safety | EFF_T3 | Summary Statistics for change from baseline PGA Scores by Treatment and Visit | | IA, SAC |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.13. | Safety | EFF_T4 | Summary of Statistical Analysis Results for Change from Baseline PGA Score by Visit | Include related estimated LSMeans and treatment differences. Footnote: | IA, SAC |
| PGA "C | Clear"/"Almost | Clear" | | | |
| 3.14. | Safety | EFF_T2 | Frequency: PGA score of Clear/Almost Clear by Treatment and Visit | Clear/Almost is a score of 0 or 1 | IA, SAC |
| 3.15. | Safety | EFF_T1 | GEE Point Estimate and 95% CI for PGA Score of Clear / Almost Clear by Visit | Footnote: | IA, SAC |
| BSA | | | | | |
| 3.16. | Safety | EFF_T3 | Summary Statistics for BSA scores by Treatment and Visit | | IA, SAC |
| 3.17. | Safety | EFF_T3 | Summary Statistics for change from baseline BSA scores by Treatment and Visit | | IA, SAC |
| 3.18. | Safety | EFF_T4 | Summary of Statistical Analysis Results for Change from Baseline BSA score by Visit | | IA, SAC |
| DLQI | | | | | |
| 3.19. | Safety | EFF_T3 | Summary Statistics for DLQI scores by Treatment and Visit | | IA, SAC |
| 3.20. | Safety | EFF_T3 | Summary Statistics for change from baseline DLQI scores by Treatment and Visit | | IA, SAC |
| 3.21. | Safety | EFF_T4 | Summary of Statistical Analysis Results for Change from Baseline DLQI score by Visit | | IA, SAC |
| VAS Ito | h Score | | | | |
| 3.22. | Safety | EFF_T3 | Summary Statistics for VAS scores by Treatment and Visit | | IA, SAC |
| 3.23. | Safety | EFF_T3 | Summary Statistics for change from baseline VAS scores by Treatment and Visit | | IA, SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.24. | Safety | EFF_T4 | Summary of Statistical Analysis Results for Change from Baseline VAS score by Visit | | IA, SAC |

# 11.13.8. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PLSS | | | | | |
| 3.1. | Safety | FE1 | Individual PLSS scores over Time by Treatment | Panel plot by subject, line colour to reflect treatment group, subjid as cell header | IA, SAC |
| 3.2. | Safety | FE2 | Mean (+/-SD) PLSS Scores over Time by Treatment | | IA, SAC |
| 3.3. | Safety | FE2 | Point Estimates and 95% CI for Change from Baseline in PLSS Score over Time by Treatment | Grey dashed ref line at y=0 | IA, SAC |
| PASI | • | | | | |
| 3.4. | Safety | FE1 | Individual PASI Scores over Time by Treatment | Panel plot by subject, line colour to reflect treatment group, subjid as cell header | IA, SAC |
| 3.5. | Safety | FE2 | Mean (+/-SD) PASI Scores over Time by Treatment | | IA, SAC |
| 3.6. | Safety | FE2 | Point Estimates and 95% CI for Change from Baseline in PASI Score over Time by Treatment | Grey dashed ref line ay y=0 | IA, SAC |
| 3.7. | Safety | FE2 | Proportion of Subjects Who Achieved PASI50 over Time by Treatment | Line graph Treatment on the same plot | IA, SAC |
| 3.8. | Safety | FE3 | Odds Ratio and 95% CI for Achieving PASI50 over Time by Treatment | | IA, SAC |
| 3.9. | Safety | FE2 | Proportion of Subjects Who Achieved PASI75 over Time by Treatment | Line graph Treatment on the same plot | IA, SAC |
| 3.10. | Safety | FE3 | Odds Ratio and 95% CI for Achieving PASI75 over Time by Treatment | | IA, SAC |
| 3.11. | Safety | FE2 | Proportion of Subjects Who Achieved PASI90 over Time by Treatment | Line graph Treatment on the same plot | IA, SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12. | Safety | FE3 | Odds Ratio and 95% CI for Achieving PASI90 over Time by Treatment | | IA, SAC |
| PGA | | | | | |
| 3.13. | Safety | FE1 | Individual PGA Scores over Time by Treatment | Panel plot by subject, line colour to reflect treatment group, subjid as cell header | IA, SAC |
| 3.14. | Safety | FE2 | Mean (+/-SD) PGA Scores over Time by Treatment | | IA, SAC |
| 3.15. | Safety | FE3 | Point Estimates and 95% CI for Change from Baseline in PGA Score over Time by Treatment | Grey dashed ref line ay y=0 | IA, SAC |
| PGA "C | Clear"/"Almost | Clear" | | | |
| 3.16. | Safety | FE2 | Proportion of Subjects Who Achieve PGA Score of Clear / Almost Clear over Time by Treatment | | IA, SAC |
| 3.17. | Safety | FE3 | Odds Ratio and 95% CI for Achieving PGA Score of Clear over Time by Treatment | | IA, SAC |
| BSA | | | | | |
| 3.18. | Safety | FE1 | Individual BSA Scores over Time by Treatment | Panel plot by subject, line colour to reflect treatment group, subjid as cell header | IA, SAC |
| 3.19. | Safety | FE2 | Mean (+/-SD) BSA Scores over Time by Treatment | | IA, SAC |
| 3.20. | Safety | FE3 | Point Estimates and 95% CI for Change from Baseline in BSA Score over Time by Treatment | Grey dashed ref line ay y=0 | IA, SAC |
| DLQI | | | | | |
| 3.21. | Safety | FE1 | Individual DLQI Scores over Time by Treatment | Panel plot by subject, line colour to reflect treatment group, subjid as cell header | IA, SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.22. | Safety | FE2 | Mean (+/-SD) DLQI Scores over Time by Treatment | | IA, SAC |
| 3.23. | Safety | FE3 | Point Estimates and 95% CI for Change from Baseline in DLQI Score over Time by Treatment | Grey dashed ref line ay y=0 | IA, SAC |
| VAS ito | h score | | | | |
| 3.24. | Safety | FE1 | Individual VAS itch Scores over Time by Treatment | Panel plot by subject, line colour to reflect treatment group | IA, SAC |
| 3.25. | Safety | FE2 | Mean (+/-SD) VAS itch Scores over Time by Treatment | | IA, SAC |
| 3.26. | Safety | FE3 | Point Estimates and 95% CI for Change from Baseline in VAS itch Score over Time by Treatment | Grey dashed ref line ay y=0 | IA, SAC |

# 11.13.9. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK con | PK concentration data | | | | |
| 4.1. | PK | PKPT1 | Summary of Plasma GSK2982772 Pharmacokinetic Concentration-Time Data (ng/mL) | | IA, SAC |
| 4.2. | PK | PKPT1 | Summary of Skin GSK2982772 Pharmacokinetic Concentration-<br>Time Data (ng/mL) | | IA, SAC |

# 11.13.10. Pharmacokinetic Figures

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| ndivid | ual concentrati | on plots | | | |
| 4.1. | PK | PKCF1P | Individual Plasma GSK2982772 Concentration-Time Plot by Subject (Linear and Semi-Log) | Page by: subject Panel: linear and semi-log x-axis: actual relative time y-axis: PK concentration Legend: Visit | IA, SAC |
| <b>vl</b> ean/n | nedian concent | ration plots | | | |
| 4.2. | PK | PKCF2 | Mean (+ SD) plot: Plasma GSK2982772 concentrations (linear and semi-log) | Panel: linear and semi-log<br>x-axis: planned relative time<br>y-axis: PK concentration<br>Legend: active treatment | IA, SAC |
| 4.3. | PK | PKCF3 | Median (range) plot: GSK2982772 Plasma concentrations (linear and semi-log) | Panel: linear and semi-log<br>x-axis: planned relative time<br>y-axis: PK concentration<br>Legend: active treatment | IA, SAC |
| ndivid | ual concentrati | on plots | | | |
| 4.4. | PK | PKCF1P | Individual Skin GSK2982772 Concentration-Time Plot by Subject (Linear and Semi-Log) | Page by: subject Panel: linear and semi-log x-axis: actual relative time y-axis: PK concentration Legend: Visit | IA, SAC |
| Mean/n | nedian concent | ration plots | | | |
| 4.5. | PK | PKCF2 | Mean (+ SD) plot: Skin GSK2982772 concentrations (linear and semi-log) | Panel: linear and semi-log x-axis: planned relative time y-axis: PK concentration Legend: active treatment | IA, SAC |
| Pharma | Pharmacokinetic : Figures | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| 4.6. | PK | PKCF3 | Median (range) plot: Skin GSK2982772 concentrations (linear and semi-log) | Panel: linear and semi-log x-axis: planned relative time y-axis: PK concentration Legend: active treatment | IA, SAC | | | |

# 11.13.11. Pharmacodynamic and / or Biomarker Tables

| Pharma | codynamic (ar | nd or Biomarker) : | Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Inflamn | natory Biomark | ers in Skin | | | |
| 5.1. | Safety | PD1 | Summary of Histopathological Scoring in Psoriatic Lesional Biopsies | By parameter / (epidermis/dermis)<br>K16: 0 or 1 | IA, SAC |
| 5.2. | Safety | PD3 | Summary of Percentage Change in Histopathological Scoring in Psoriatic Lesional Biopsies | | IA, SAC |
| 5.3. | Safety | EFF_T4 | Adjusted Mean (95% CI) Percentage Change in Histopathological Scoring of Psoriatic Lesional Biopsy | Present %CVb instead of SE | IA, SAC |
| mRNA i | in Skin | | | | |
| 5.4. | Safety | PD2 | Summary of mRNA Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies | | IA, SAC |
| 5.5. | Safety | PD_T2 | Frequency Table Summarising the Number of Probe Sets with Various Fold Change in Psoriatic Lesional Biopsies | Use cut-offs 1.5 and -1.5 initially.<br>Change to -1.25 and 1.5 if no one<br>achieves the initial cut-offs | IA, SAC |
| 5.6. | Safety | PD_T3 | Summary of Adjusted Mean Fold Changes in mRNA Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies | If Adj Mean FC lies between -1 and 1 then do not include on table | IA, SAC |
| Inflami | matory Biomar | kers in Blood | | | |
| 5.7. | Safety | PD1 | Summary Statistics of Blood Inflammatory Biomarkers | One page for each cell type/measure by visit/time and treatment | IA, SAC |
| 5.8. | Safety | PD2 | Summary of Percentage Change in Blood Inflammatory Biomarkers | One page for each cell type/measure by visit/time and treatment | IA, SAC |
| 5.9. | Safety | EFF_T4 | Adjusted Mean (95% CI) Percentage Change in Blood Inflammatory Biomarkers | Present %CVb instead of SE | IA, SAC |
| Pathwa | y and Target E | ngagement | | | |

| Pharma | Pharmacodynamic (and or Biomarker) : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.10. | Safety | | Summary of TEAR1 % Target Engagement in Blood | % Target Engagement by visit/time,<br>Refer to 200975/Partb_final for display | IA, SAC |
| 5.11. | Safety | | Adjusted Mean (95% CI) TEAR1 % Target Engagement in Blood | Refer to 200975/Partb_final for display | IA, SAC |
| 5.12. | Safety | | Summary of TEAR1 % Target Engagement in Skin | % Target Engagement by visit/time,<br>Refer to 200975/Partb_final for<br>display | IA, SAC |
| 5.13. | Safety | | Adjusted Mean (95% CI) TEAR1 % Target Engagement in Skin | Refer to 200975/Partb_final for display | IA, SAC |

# 11.13.12. Pharmacodynamic (and / or Biomarker) Figures

| Pharma | acodynamic (ar | nd or Biomarker) : | Figures | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Inflamr | natory Biomark | ers in Skin | | | |
| 5.14. | Safety | FE1 | Individual Subject Profiles for Histopathological Scoring in Psoriatic Lesional Biopsies | Page by biomarker and location (dermis/epidermis) Panel plot, line colours by treatment group, subjid as cell header | IA, SAC |
| 5.15. | Safety | FE2 | Adjusted Mean (95% CI) Percentage Change in Histopathological Scoring of Psoriatic Lesional Biopsy | Reference line at y=0, grey dashed style | IA, SAC |
| mRNA | in Skin | | | | |
| 5.16. | Safety | FE1 | Individual Subject Profiles for mRNA Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies | Panel plot, line colours by treatment group, subjid as cell header | IA, SAC |
| 5.17. | Safety | FE4 | Adjusted Mean Intensities for for mRNA Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies | Y xais – log2 scale | IA, SAC |
| 5.18. | Safety | FE5 | Adjusted Mean (95% CI) Fold Change in mRNA Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies | If Adj Mean FC lies between -1 and 1 then do not include on table Include band from FC -1 to 1, transparency 0.5 | IA, SAC |
| Inflam | matory Biomar | kers in Blood | | | |
| 5.19. | Safety | FE1 | Summary Statistics of Blood Inflammatory Biomarkers | Page by biomarker Panel plot, line colours by treatment group, subjid as cell header | IA, SAC |
| 5.20. | Safety | FE2 | Adjusted Mean (95% CI) Percentage Change in Blood Inflammatory Biomarkers | Reference line at y=0, grey dashed style | IA, SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Program | nming No | otes | | Deliverable<br>[Priority] |
|---|---|---|---|---|---|---|---|---|
| Pathwa | y and Target E | ngagement | | | | | | |
| 5.21. | Safety | FE1 | Individual Subject Profiles for TEAR1 % Target Engagement in Blood | | t, line colo<br>bjid as cell | | atment | IA, SAC |
| 5.22. | Safety | FE2 | Adjusted Mean (95% CI) TEAR1 % Target Engagement in Blood | | | | | IA, SAC |
| 5.23. | Safety | FE1 | Individual Subject Profiles for TEAR1 % Target Engagement in Skin | | t, line colo<br>bjid as cell | | atment | IA, SAC |
| 5.24. | Safety | FE2 | Adjusted Mean (95% CI) TEAR1 % Target Engagement in Skin | | | | | IA, SAC |
| 5.25. | Safety | FE6 | Scatter Plot of TEAR 1 % Target Engagement in Blood vs. | Include be<br>percentile<br>ref line at | | wer 10 <sup>th</sup> a<br>PD, and gro | | IA, SAC |
| 0.20. | | TEAR1 % Target Engagement in Skin by Treatment Group | TEAR1 % Target Engagement in Skin by Treatment Group | | percen<br>tile | n | Perce<br>ntile | , |
| | | | | Blood | 85.3% | 95% | 98.4% | |
| | | | | Skin | 70.3% | 88.5% | 96.1<br>% | |

| Pharma | Pharmacodynamic (and or Biomarker) : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.26. | Safety | FE7 | Scatter Plot of TEAR1 % Target Engagement in Skin vs. Percentage Change in Histopathological Scoring in Psoriatic Lesional Biopsies | Page by biomarker and location (dermis/epidermis) X axis – TE Skin, y axis - % Chg Biomarker Markers by treatment group | IA, SAC |
| 5.27. | Safety | FE7 | Scatter Plot of TEAR1 % Target Engagement in Skin vs. Fold Change in mRNA Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies | Page by biomarker and location (dermis/epidermis) X axis – TE Skin, y axis - % Chg Biomarker Markers by treatment group Band for FC between -1 to 1 | IA, SAC |

# 11.13.13. Biomarker / Efficacy Figures

| Pharma | acodynamic (ar | nd or Biomarker) : | Figures | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.28. | Safety | FE7 | Scatter Plot of TEAR1 % Target Engagement in Skin vs. Percentage Change in PLSS | Page by biomarker and location (dermis/epidermis) X axis – TE Skin, y axis - % Chg Biomarker Markers by treatment group Band for FC between -1 to 1 | IA, SAC |
| 5.29. | Safety | FE7 | Scatter Plot of TEAR1 % Target Engagement in Skin vs. Percentage Change in PASI | Page by biomarker and location (dermis/epidermis) X axis – TE Skin, y axis - % Chg Biomarker Markers by treatment group Band for FC between -1 to 1 | IA, SAC |

# 11.13.14. ICH Listings

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | misation | | | | |
| 1. | Safety | CP_TA1 | Listings of Randomised and Actual Treatments | | IA, SAC |
| Subjec | t Disposition | | | | |
| 2. | All subjects | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | IA, SAC |
| 3. | Safety | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | IA, SAC |
| 4. | Safety | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | ICH E3 | IA, SAC |
| 5. | Safety | TA1 | Listing of Planned and Actual Treatments | IDSL | IA, SAC |
| Protoc | ol Deviations | | | | |
| 6. | Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 Listing also includes analysis population exclusions. | IA, SAC |
| 7. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | IA, SAC |
| Popula | tion Analysed | | | | |
| 8. | All Subjects | SA3a | Listing of Subjects Excluded from Any Population | ICH E3 e.g., subjects screened but not randomized, subjects randomized but not treated, subjects with deviations leading to exclusion from per protocol population (can be separate listing per population). | IA, SAC |

| Demog | raphic and Bas | seline Characteris | tics | | |
|---|---|---|---|---|---|
| 9. | Safety | DM2 | Listing of Demographic Characteristics | ICH E3 | IA, SAC |
| 10. | Safety | DM9 | Listing of Race | ICH E3 | IA, SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | Safety | CP_CM3 | Listing of Concomitant Medications | IDSL | IA, SAC |
| Exposu | re and Treatmo | ent Compliance | | | • |
| 12. | Safety | EX3 | Listing of Exposure Data | ICH E3 | IA, SAC |
| Advers | e Events | | | | |
| 13. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | IA, SAC |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | IA, SAC |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | IA, SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | • |
| 16. | Safety | CP_AE8a | Listing of Serious Adverse events | ICH E3 | IA, SAC |
| 17. | Safety | SAE Reasons | Listing of Reasons for Considering as a Serious Adverse Event | FDA Note: IDSL shell in development. | IA, SAC |
| 18. | Safety | CP_AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | IA, SAC |
| Hepato | biliary (Liver) | | | | |
| 19. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | IDSL | IA, SAC |
| 20. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | IDSL | IA, SAC |

| All Labo | oratory | | | | |
|---|---|---|---|---|---|
| 21. | Safety | LB5 | Listing of Laboratory Data for Subjects with Abnormalities of Potential Clinical Concern | ICH E3 Include fasted or non-fasted. Include subjects that have both absolute and change from baseline PCI | IA, SAC |
| 22. | Safety | LB5 / LB6 | Listing of Laboratory Data Abnormalities of Potential Clinical Importance | Include fasted or non-fasted. | IA, SAC |
| ECG | | | | | |
| 23. | Safety | CP_EG3 | Listing of All ECG Values for Subjects with a Value of Potential Clinical Importance | IDSL Include absolute PCI subjects. Footnote: H=High absolute, L= Low absolute." | IA, SAC |
| 24. | Safety | CP_EG3 | Listing of All ECG Changes for Subjects with a Value of Potential Clinical Importance | IDSL Include change from baseline PCI subjects. Footnote: H=High change from baseline value, L= Low change from baseline value | IA, SAC |
| 25. | Safety | CP_EG3 | Listing of ECG Values of Potential Clinical Importance | "Include absolute PCIs. Footnote: H=High absolute, L= Low absolute." | IA, SAC |
| 26. | Safety | CP_EG3 | Listing of ECG Changes of Potential Clinical Importance | "Include change from baseline PCIs. Footnote: H=High change, L= Low changee." | IA, SAC |
| 27. | Safety | CP_EG5 | Listing of Abnormal ECG Findings | IDSL | IA, SAC |
| Vital Sig | gns | | | | |

| 28. | Safety | CP_VS4 | Listing of All Vital Signs for Subjects with Values of Potential Clinical Importance | "Include both absolute and change from baseline PCI subjects. Footnote: H=High, L=Low H1=Lower Increase, H2=Upper Increase, L1=Lower Decrease, L2=Upper Decrease" | IA, SAC |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

# 11.13.15. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Colum | bia Suicide Sev | erity Rating Scale | (C-SSRS) | • | |
| 29. | Safety | ECSSRS4 | Listing of C-SSRS suicidal Ideation and Behaviour Data | | IA, SAC |
| 30. | Safety | ECSSRS5 | Listing of C-SSRS Suicidal Behaviour Details | | IA, SAC |
| Pharma | acokinetic | | | | |
| 31. | PK | PKCL1X | Listing of Blood GSK2982772 Pharmacokinetic Concentration-<br>Time (ng/mL) Data | | IA, SAC |
| 32. | PK | PKCL1X | Listing of Skin GSK2982772 Pharmacokinetic Concentration-<br>Time (ng/mL) Data | | IA, SAC |
| Pharma | acodynamic | | | | |
| 33. | Safety | LS2 | Listing of Histopathological Scoring in Psoriatic Lesional Biopsies | Including, but not limited to K16, CD3/Cd11c, CD161, elastase positive dermal cells and epidermal thickness. | IA, SAC |
| 34. | Safety | LS1 | Listing of mRNA Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies | Including, but not limited to CRP, VEGF, S100A8, S100A9, IL-17, IL-22 and TNF. | IA, SAC |
| 35. | Safety | LS2 | Listing of Blood Inflammatory Biomarkers | | IA, SAC |
| 36. | Safety | | Listings of TEAR1 % Target Engagement | See 200975/partb_final | IA, SAC |
| 37. | Safety | n/a | Raw SAS Output of Statistical Analysis of Histopathological Scoring in Psoriatic Lesional Biopsies | | IA, SAC |
| 38. | Safety | n/a | Raw SAS Output of Statistical Analysis of Inflammatory Gene<br>Transcripts in Psoriatic Lesional Biopsies | | IA, SAC |
| 39. | Safety | n/a | Raw SAS Output of Statistical Analysis of Blood Inflammatory Biomarkers | | IA, SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 40. | Safety | n/a | Raw SAS Output of Statistical Analysis of TEAR1 % Target Engagement | | IA, SAC |
| Efficac | y | | | | |
| 41. | Safety | LS2 | Listings of PLSS absolute and change from baseline score | | IA, SAC |
| 42. | Safety | LS2 | Listings of PASI absolute, change from baseline, percentage change from baseline, PASI50, PASI75 and PASI90 status | | IA, SAC |
| 43. | Safety | LS2 | Listing of PGA categories by treatment over time | | IA, SAC |
| 44. | Safety | LS2 | Listing of BSA absolute and change from baseline score | | IA, SAC |
| 45. | Safety | LS2 | Listing of DLQI Absolute and Change From Baseline Score | | IA, SAC |
| 46. | Safety | LS2 | Listings of VAS Absolute and Change From Baseline Score | | IA, SAC |
| 47. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for<br>Percentage Change From Baseline PLSS Score | | IA, SAC |
| 48. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for Change From Baseline PASI Score | | IA, SAC |
| 49. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for PASI50 Score | | IA, SAC |
| 50. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for PASI75 Score | | IA, SAC |
| 51. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for PASI90 Score | | IA, SAC |
| 52. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for Change from Baseline PGA Score | | IA, SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 53. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for PGA Score of Clear / Almost Clear | | IA, SAC |
| 54. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for Change From Baseline BSA score | | IA, SAC |
| 55. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for Change From Baseline BSA score | | IA, SAC |
| 56. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for Change From Baseline DLQI score | | IA, SAC |
| 57. | Safety | n/a | RAW SAS Output of Statistical Analysis Results for Change From Baseline VAS score | | IA, SAC |

# 11.14. Appendix 14: Example Mock Shells for Data Displays

203167

Example : LS1 Page 1 of n

Protocol : 203167
Population : Safety

Listing XX:

Listing of Absolute, Percentage Inhibition and Maximum Percentage Inhibition in qPCR Expression

| Gene | Treatment | Subject | Visit | CT1/CT2/<br>CTAVG/<br>Copy<br>Number | Value | Percentage<br>Inhibition<br>[1] | Maximum<br>Percentage<br>Inhibition<br>[2] |
|---|---|---|---|---|---|---|---|
| XXXXGENE | GSKXXXXXX XXmg | xxxx | Screening | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX<br>XX.XXX | | |
| | | | Baseline | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX<br>XX.XXX | x.xxx | |
| | | | Week X | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX | x.xxx | |

203167

Example : LS2 Page 1 of n

Protocol : 203167
Population : Safety

Listing XX:

Listing of Raw, Change from baseline and Percent Change in [variable]

| Treatment | Subject | Visit | Visit<br>date | Study<br>day | Histopatholgical<br>Scoring | Raw | Change | Percent<br>Change |
|---|---|---|---|---|---|---|---|---|
| Placebo | xxx | xxx | XX/XX/XX | Day 1 | K16<br>CD3/CD11c<br>CD161<br>Elactase +ve cels<br>epidermal thickness | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X | , | |
| | | XXX | XX/XX/XX | Day 43 | K16<br>CD3/CD11c<br>CD161<br>Elactase +ve cels<br>epidermal thickness | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X | XXX.X<br>XXX.X<br>XXX.X<br>XXX.X |

203167

Example EFF T1 

Protocol: 203167 Population: Safety

Table XX: GEE Point Estimate and 95% CI for PASIXX by Week

| Comparison | Parameter | Odds Ratio | Odds Ratio |
|---|---|---|---|
| GSK2982772 vs Placebo<br>GSK2982772 vs Placebo<br>GSK2982772 vs Placebo | PASIXX at Day 1 PASIXX at Day 15 PASIXX at Day 29 | x.xx<br>x.xx<br>x.xx | (x.xx, x.xx)<br>(x.xx, x.xx)<br>(x.xx, x.xx) |

Example EFF T2

Protocol: 203167 Population: Safety


Table XX: Frequency Table for PASI50, PASI75 by week

| | | Placebo | 100mg | 200mg | 400mg |
|-----------|--------|----------|---------|---------|---------|
| | | 1 140000 | roomg | Zoomg | Toomig |
| Parameter | Visit | N=x | N=x | N=x | N =x |
| PASI50 | Day 1 | nn/nn | nn / nn | nn / nn | nn / nn |
| | | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| | Day 15 | nn / nn | nn / nn | nn / nn | nn / nn |
| | | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| | Day 29 | nn / nn | nn / nn | nn / nn | nn / nn |
| | | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| PASI75 | Day 1 | nn / nn | nn / nn | nn / nn | nn / nn |
| | | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| | Day 15 | nn / nn | nn / nn | nn / nn | nn / nn |
| | | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| | Day 29 | nn / nn | nn / nn | nn / nn | nn / nn |
| | | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| PASI90 | Day 1 | nn / nn | nn / nn | nn / nn | nn / nn |
| | • | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| | Day 15 | nn / nn | nn / nn | nn / nn | nn / nn |
| | - | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| | Day 29 | nn / nn | nn / nn | nn / nn | nn / nn |
| | - | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |

203167

Example EFF\_T3 

Protocol: 203167
Population: Safety

Table XX: Summary Statistics (Mean +/- SD) for Actual and Change from Baseline [Continuous Parameter] by Treatment and Week

| Parameter | Treatment | N | Visit | n | Mean | {95% CI<br>(Lower,Upper)} | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| Continuous | GSK2982772 | 18 | Day 1 | 18 | XXXX.XX | (xxxx.xx,xxxxxx) | XX.XXX | XXXX.XX | XXXX.X | XXXX.X |
| Parameter | | | Day 15 | 18 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | xxxx.xx | XXXX.X | XXXX.X |
| | | | Day 29 | 18 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XX | xxxx.xx | XXXX.X | XXXX.X |
| | Placebo | 6 | Day 1 | 6 | xxxx.xx | (xxxx.xx,xxxxx) | XX.XXX | xxxx.xx | xxxx.x | xxxx.x |
| | | | Day 15 | 6 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | xxxx.xx | XXXX.X | xxxx.x |
| | | | Day 29 | 6 | XXXX.XX | (xxxx.xx,xxxxxx) | XX.XXX | xxxxx | XXXX.X | XXXX.X |


Example: EFF\_T4
Protocol: 203167

Population: Safety

Table x.x:

Repeated Measures Analysis of the Change from Baseline in [Continuous Parameter] at Each Visit

| Visit | Treatment<br>Group | n | LSMean | Standard<br>Error | 95% CI for<br>LS Mean | Differen<br>from<br>Placebo | ce 95% CI for<br>Difference<br>(Lower, Upper) |
|---|---|---|---|---|---|---|---|
| Week 1 | Placebo<br>GSK2982772 | X<br>X | x.xx<br>x.xx | x.xxx<br>x.xxx | (x.xx, x.xx) | x.xx | (x.xx, x.xx) |
| Week 2 | Placebo<br>GSK2982772 | x | x.xx<br>x.xx | x.xxx<br>x.xxx | (x.xx, x.xx)<br>(x.xx, x.xx) | x.xx | (x.xx, x.xx) |

Repeated Measures Analysis adjusted for Baseline Score, Treatment Group, Visit and Treatment Group by Visit Interaction

Example: PD\_T1
Protocol: 203167

tocol:  $2\overline{0}3167$  Page 1 of x

Population: Safety

### Listing XX:

Listing of Absolute, Percentage Inhibition and Maximum Percentage Inhibition in mRNA Expression

| Gene | Treatment | Subject | Visit | CT1/CT2/<br>CTAVG/<br>Copy<br>Number | Value | Percentage<br>Inhibition<br>[1] | Maximum<br>Percentage<br>Inhibition<br>[2] |
|---|---|---|---|---|---|---|---|
| XXXXGENE | GSKXXXXXX XXmg | xxxx | Screening | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX<br>XX.XXX | | |
| | | | Baseline | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX<br>XX.XXX | x.xxx | |
| | | | Week X | CT1<br>CT2<br>CTAVG<br>NORMALISED | XX.XXX<br>XX.XXX<br>XX.XXX | x.xxx | |


Example: PD\_T2
Protocol: 203167

Population: Safety

Table XX.XX :

Frequency table summarising the number of probe sets in various fold change Fold Change

| Probeset | Gene | Visit | N | n | Treatment | < | 1.5 | >1 | .5 |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | Baseline | XX | XX | Placebo<br>GSKXXXXXX XXmg | | (xx.xx)<br>(xx.xx) | | (xx.xx)<br>(xx.xx) |
| | | WEEK xx | XX | XX | Placebo<br>GSKXXXXXX XXmg | | (xx.xx)<br>(xx.xx) | | (xx.xx)<br>(xx.xx) |
| | | WEEK xx | XX | XX | Placebo<br>GSKXXXXXX XXmg | | (xx.xx)<br>(xx.xx) | | (xx.xx)<br>(xx.xx) |

Example: PD\_T3
Protocol: 203167
Population: Safety

Protocol: 203167 Page 1 of x

| Treatment<br>Group | n<br>Adjusted Mean<br>95% CI | n<br>Adjusted Mean<br>95% CI | Fold Chg. From<br>Baseline<br>95% CI | Comparison to Placebo<br>Fold Change<br>95% CI |
|---|---|---|---|---|
| Placebo S | 4 | 4 | | |
| D/RD (4W) | 10033.48 | 13337.45 | 1.33 | |
| (N=6) | (5015.87, 20070.45) | (4806.65, 37008.63) | (-1.24, 2.19) | |
| GSK 60mg B | ID 8118.18 | 6830.11 | -1.19 | -1.58 |
| (N=4) | (3264.70, 20187.10) | (2150.27, 21695.19) | (-1.96, 1.39) | (-3.21, 1.28) |
| GSK 60mg T | ID 9 | 9 | | |
| 15mg/kg | 6459.95 | 6471.40 | 1.00 | -1.33 |
| (N=15) | (3943.96, 10580.99) | (3139.22, 13340.56) | (-1.42, 1.43) | (-2.45, 1.39) |

203167

Example: FE1 

Protocol: 203167
Population: Safety

Table X

Individual [Continuous Parameter] Scores over Time by Treatment



USER ID:directory/program.sas 01JAN2002 12:01

Example: FE2
Protocol: 203167
Population: Safety




203167


Example: FE3
Protocol: 203167

Protocol: 203167
Population: Safety

Table X
Treatment Difference and 95% CI of [Continuous Parameter]



Example: FE4
Protocol: 203167
Population: Safety


Figure XX.XX: Adjusted mean probe set intensity values (95% CI) by time from xxxx

Gene ID: XXXX




Example: FE5
Protocol: 203167

Population: Safety

Figure XX.XX: Adjusted Fold Change in mRNA Expression

Gene ID: XXXX



Example: FE6
Protocol: 203167
Population: Safety


Figure XX.XX:


## Plasma TE vs Skin TE



Example: FE7
Protocol: 203167

Population: Safety

Figure XX.XX: Skin TE vs Effiacy/Biomarkers

